CLINICAL TRIAL: NCT01243424
Title: A Multicentre, International, Randomised, Parallel Group, Double Blind Study to Evaluate Cardiovascular Safety of Linagliptin Versus Glimepiride in Patients With Type 2 Diabetes Mellitus at High Cardiovascular Risk.
Brief Title: CAROLINA: Cardiovascular Outcome Study of Linagliptin Versus Glimepiride in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.74; 2009-013157-15 (EudraCT Number)
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Results first posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- linagliptin (Experimental): patient to receive linagliptin or glimepiride placebo over encapsulated tablet Quaque die (QD)
  Interventions: Drug: linagliptin; Drug: glimepiride placebo
- glimepiride 1-4 mg QD (Active Comparator): patient to receive glimepiride 1-4 mg or linagliptin placebo tablet Quaque die (QD)
  Interventions: Drug: glimepiride; Drug: linagliptin placebo

INTERVENTIONS:
Drug: linagliptin — linagliptin tablets 5mg QD
  Arms: linagliptin
Drug: glimepiride — glimepiride over-encapsulated tablet 1-4 mg QD
  Arms: glimepiride 1-4 mg QD
Drug: linagliptin placebo — linagliptin placebo
  Arms: glimepiride 1-4 mg QD
Drug: glimepiride placebo — glimepiride placebo
  Arms: linagliptin

SUMMARY:
The aim of the study is to investigate the longterm impact on cardiovascular morbidity and mortality, relevant efficacy parameters (e.g., glycaemic parameters) and safety (e.g., weight and hypoglycaemia) of treatment with linagliptin in patients with type 2 diabetes at elevated cardiovascular risk receiving usual care, and compare outcome against glimepiride.

ELIGIBILITY:
Inclusion criteria:

1. Type 2 diabetes
2. Elevated glycosylated haemoglobin (HbA1c): 6.5 - 8.5%, inclusive, if treatment naïve or mono-/dual therapy with metformin and/or an alpha-glucosidase inhibitor; 6.5 - 7.5%, inclusive, if treatment with sulphonylurea/glinide in mono- or dual (with metformin OR an alpha-glucosidase inhibitor) therapy)
3. Pre-existing cardiovascular disease OR specified diabetes end-organ damage OR age => 70 years OR two or more specified cardiovascular risk factor
4. BMI =< 45kg/m²
5. age between >= 40 and =< 85 years
6. signed and dated written International Conference of Harmonisation( ICF)
7. stable anti-diabetic background for at least 8 wks before study start

Exclusion criteria:

1. Type 1 diabetes
2. Treatment with other antidiabetic drugs (e.g. rosiglitazone, pioglitazone, Glucagon-like peptide 1 (GLP-1) analogue/agonists, Dipeptidyl-peptidase IV (DPP-IV) inhibitors or any insulin) prior to informed consent (previous short term use of insulin (up to two weeks) is allowed if taken at least 8 weeks prior informed consent)
3. treatment with any anti-obesity drug less than 3 months before ICF
4. uncontrolled hyperglycemia
5. previous or planned bariatric surgery or intervention
6. current or planned system corticoid treatment
7. change in thyroid hormones treatment
8. acute liver disease or impaired hepatic function
9. pre-planned coronary artery revascularization within 6 months of ICF
10. known hypersensitivity to any of the components
11. Inappropriateness of glimepiride treatment for renal safety issues according to local prescribing information
12. congestive heart failure class III or IV
13. acute or chronic metabolic acidosis
14. hereditary galactose intolerance
15. alcohol or drug abuse
16. participation in another trail with IMP given 2 months before Investigational Medicinal/Medical Product (IMP) start
17. pre-menopausal women who are nursing or pregnant or of child-bearing potential and not willing to use acceptable method of birth control
18. patients considered reliable by the investigator
19. acute coronary syndrome =< 6 wks before ICF
20. stroke or Transient Ischemic Attack (TIA) =< 3 months prior to ICF

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6103 (Actual)
Dates: Start 2010-11-11 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (611):
- United States (175):
  - North Alabama Research Center, LLC, Athens, Alabama
  - Alabama Internal Medicine, PC, Birmingham, Alabama
  - Cahaba Research, Inc., Birmingham, Alabama
  - Internal Medicine Center, LLC, Mobile, Alabama
  - Diagnostic and Medical Clinic, Mobile, Alabama
  - Extended Arm Physicians, Inc., Montgomery, Alabama
  - Office of Dr. Terence T. Hart MD, Tuscumbia, Alabama
  - Advanced Clinical Research, Pell City, Alaska
  - Clinical Research Advantage, Inc./Rita B. Chuang, MD, LLC, Mesa, Arizona
  - Genova Clinical Research, Tucson, Arizona
  - Quality of Life Medical & Research Center, Tucson, Arizona
  - Northeast Arkansas Baptist Clinic, Jonesboro, Arkansas
  - Medical Investigations, Inc, Little Rock, Arkansas
  - Aureus Research, Inc, Little Rock, Arkansas
  - Desert Oasis Healthcare, Bermuda Dunes, California
  - Edinger Medical Group and Research Center, Fountain Valley, California
  - Clinical Trials of St. Jude Heritage Med. Group, Fullerton, California
  - Long Beach Center for Clinical Research, Long Beach, California
  - Office of Dr. Richard S. Cherlin, Los Gatos, California
  - Providence Clinical Research, North Hollywood, California
  - Chaparral Medical Group, Inc, Pomona, California
  - ARI Clinical Trials, Inc, Redondo Beach, California
  - San Diego Sports Medicine and Family Health Center, San Diego, California
  - West Coast Research, LLC, San Ramon, California
  - University of California Los Angeles, Sylmar, California
  - Metabolic Institute of America, Tarzana, California
  - Matrix Research Institute, Tustin, California
  - Orange County Research Center, Tustin, California
  - Westlake Medical Research, Westlake Village, California
  - Clinical Research Advantage, Inc./Rita B. Chuang, MD, LLC, Colorado Springs, Colorado
  - East Coast Medical Associates, Boca Raton, Florida
  - Todd Kazdan, DO Family Practice, Davie, Florida
  - Century Clinical Research, Inc, Daytona Beach, Florida
  - Doral Research Center, Doral, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - Alan Graff, MD, PA, Fort Lauderdale, Florida
  - M & O Clinical Research, LLC, Fort Lauderdale, Florida
  - Eastern Research, Hialeah, Florida
  - Research in Miami Inc, Hialeah, Florida
  - Jacksonville Impotence Treatment Center, Jacksonville, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Care Partners Clinical Research LLC, Jacksonville, Florida
  - Precision Clinical Research, LLC, Lauderdale Lakes, Florida
  - Veritas Research Corporation, Miami, Florida
  - APF Research, LLC, Miami, Florida
  - Swiss Medical Research, Miami, Florida
  - University of Miami, Miami, Florida
  - South Miami Clinical Research, Miami, Florida
  - Well Pharma Medical Research, Miami, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - AppleMed Research Group, LLC, Miami, Florida
  - Kendall South Medical Center, Inc, Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Advanced Research Institute, Inc, New Port Richey, Florida
  - Sunshine Research Center, Opa-locka, Florida
  - Diabetes and Endocrine Center of Orlando, Orlando, Florida
  - Suncoast Clinical Research, Palm Harbor, Florida
  - Misal Khan, MD FRCS, ED, PA, Panama City, Florida
  - Iconic Clinical Trials, Pembroke Pines, Florida
  - Gulf Region Clinical Research Institute, Pensacola, Florida
  - St. John's Center for Clinical Research, Ponte Vedra Beach, Florida
  - Metabolic Research Institute, West Palm Beach, Florida
  - PMI Health Research Group, Atlanta, Georgia
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Albert F. Johary MD, PC, Dunwoody, Georgia
  - Georgia Clinical Research, LLC, Snellville, Georgia
  - Hayden Lake Family Physicians, Hayden Lake, Idaho
  - Boise Kidney and Hypertension Institute, Meridian, Idaho
  - Suburban Clinical Research, Bolingbrook, Illinois
  - Cedar-Crosse Research Center, Chicago, Illinois
  - John H. Stroger Jr. Hospital of Cook Country, Chicago, Illinois
  - Apex Medical Research, Chicago, Illinois
  - Pharmakon Inc, Evergreen Park, Illinois
  - American Health Network, Avon, Indiana
  - Investigators Research Group, LLC, Brownsburg, Indiana
  - American Health Network of Indiana, LLC, Franklin, Indiana
  - Mapleton Medical Center, Indianapolis, Indiana
  - American Health Network, LLC, Indianapolis, Indiana
  - McKinley Research, LLC, Mishawaka, Indiana
  - American Health Network of Indiana, LLC, Muncie, Indiana
  - MCM Clinical Research, LLC, Florence, Kentucky
  - Kentucky Diabetes Endocrinology Center, Lexington, Kentucky
  - Four Rivers Clinical Research, Inc, Paducah, Kentucky
  - Crescent City Clinical Research, Metairie, Louisiana
  - Acadia Clinical Research, LLC, Bangor, Maine
  - Office of Dr. Stephen R. Smith, MD, Baltimore, Maryland
  - Endocrine and Metabolic Consultants, Rockville, Maryland
  - Tristan Medical Enterprises, PC dba Regeneris, North Attleboro, Massachusetts
  - ClinSite, LLC, Canton, Michigan
  - Apex Medical Research, AMR Inc, Flint, Michigan
  - Westside Family Medical Center, PC, Kalamazoo, Michigan
  - Tri City Medical Centers, PC, Livonia, Michigan
  - KMED Research, Saint Clair Shores, Michigan
  - Tri-County Research, Inc, Sterling Heights, Michigan
  - Medical Research Associates, Traverse City, Michigan
  - Oakland Medical Research Center, Troy, Michigan
  - Park Nicollet Institute, Minneapolis, Minnesota
  - The Center for Clinical Trials, Inc., Biloxi, Mississippi
  - Mercy Health Research, St Louis, Missouri
  - Quality Clinical Research, Omaha, Nebraska
  - Clinical Research Advantage, Inc./Rita B. Chuang, MD, LLC, Henderson, Nevada
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Palm Medical Research Center, Las Vegas, Nevada
  - Atco Medical Associates, PC, Atco, New Jersey
  - Summit Medical Group, Clifton, New Jersey
  - USMA Clinical Research, Elizabeth, New Jersey
  - Central Jersey Medical Research, Elizabeth, New Jersey
  - Albany Medical Center / Albany Medical College, Albany, New York
  - Endocrine Associates of Long Island, PC, Smithtown, New York
  - Southgate Medical Group/ Southgate Medical Park, West Seneca, New York
  - OnSite Clinical Solutions, LLC, Asheville, North Carolina
  - Kernodle Clinic West, Burlington, North Carolina
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Internal Medicine Research, Charlotte, North Carolina
  - Gaffney Health Services, Charlotte, North Carolina
  - Durham Internal Medicine Associates, Durham, North Carolina
  - Sentara Family Medicine, Elizabeth City, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - Carolina Research Center, Inc, Shelby, North Carolina
  - Piedmont Healthcare, Statesville, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Community Health Care of Manchester, Akron, Ohio
  - Community Medical Associates, LLC, Austintown, Ohio
  - Harrison Community Research Center, Cadiz, Ohio
  - Medical Frontiers, LLC, Carlisle, Ohio
  - Genoa Medical Center, Genoa, Ohio
  - Office of Dr. Craig S. Thompson, MD, LLC, Marion, Ohio
  - RAS Health Limited, Marion, Ohio
  - Advanced Medical Research, LLC, Maumee, Ohio
  - Pharmacotherapy Research Associates, Inc, Zanesville, Ohio
  - Infinity Research Group, LLC, Oklahoma City, Oklahoma
  - Castlerock Clinical Research Consultants, LLC, Tulsa, Oklahoma
  - Oregon Medical Group, Eugene, Oregon
  - Harleysville Medical Associates, Harleysville, Pennsylvania
  - Detweiler Family Medicine & Associates, PC, Lansdale, Pennsylvania
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - Warminster Medical Associates, PC, Warminster, Pennsylvania
  - New England Center for Clinical Research, Inc, Cranston, Rhode Island
  - Hartwell Research Group, LLC, Anderson, South Carolina
  - Paris View Family Practice, Greenville, South Carolina
  - Mountain View Clinical Research, Greer, South Carolina
  - South Carolina Nephrology and Hypertension Center, Inc, Orangeburg, South Carolina
  - Carolina Diabetes & Kidney Center, Sumter, South Carolina
  - PMG Research of Bristol, Bristol, Tennessee
  - University Diabetes and Endocrine Consultants, Chattanooga, Tennessee
  - University of Tennessee, Memphis, Tennessee
  - Trinity Clinical Research, LLC, Tullahoma, Tennessee
  - KRK Medical Research, Arlington, Texas
  - Austin Center for Clinical Research, Austin, Texas
  - Punzi Medical Center, Carrollton, Texas
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - Baylor Endocrine Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Jacon Medical Research Associates, LLC, Houston, Texas
  - JVC Family Medicine, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Endocrine and Psychiastry Center, Houston, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Midland Clinical Research Center, Midland, Texas
  - Hill Country Medical Associates, New Braunfels, Texas
  - Naidu Clinic, Odessa, Texas
  - The Methodist Hospital d/b/a HMRI CCAT at Pearland, Pearland, Texas
  - Village Health Partners, Plano, Texas
  - Sun Research Institute, San Antonio, Texas
  - Northeast Clinical Research of San Antonio, LLC, Schertz, Texas
  - Kenneth Otah and Associates, Sugar Land, Texas
  - PHS Clinical Trials, Midvale, Utah
  - Highland Clinical Research, Salt Lake City, Utah
  - Burke Internal Medicine and Research, Burke, Virginia
  - Ettrick Health Center, Ettrick, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Richmond Family Practice, Richmond, Virginia
  - Larry D Stonesifer, MD Inc., PS, Federal Way, Washington
  - Premier Clinical Research, Spokane, Washington
- Argentina (16):
  - Instituto de Investigaciones Clínicas de Bahía Blanca, Bahía Blanca
  - CIPREC, CABA
  - CENUDIAB, CABA
  - Instituto Médico Especializado, Capital Federal
  - Consultorios Asociados de Endocrinología e Invest Clínica, Capital Federal
  - Instituto Cardiovascular de Corrientes Juana Francisca Cabra, Corrientes
  - Ilaim-Ceom, Córdoba
  - IPAC - Clínica Privada Caraffa SRL, Córdoba
  - Hospital Italiano de La Plata, La Plata
  - CIPADI, Mendoza
  - Instituto de Investigaciones Clinicas de Rosario, Rosario
  - Instituto de Hematología y Medicina Clínica Dr. Rubén Davoli, Rosario
  - Hospital San Bernardo, Salta
  - Investigaciones Clinicas Tucuman, San Miguel de Tucumán
  - Instituto de Investigaciones Biomédicas, Santa Fe
  - Centro de Investigaciones Clínicas del Litoral, Santa Fe
- Australia (5):
  - Royal Brisbane & Women's Hospital-Endocrinology, Herston, Queensland
  - Logan Hospital, Meadowbrook, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Eastern Clinical Research Unit, East Ringwood, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Belgium (14):
  - Blankenberge - PRAC Vileyn, Geert, Blankenberge
  - Bonheiden - HOSP Imelda, Bonheiden
  - De Pinte - PRAC Hollanders, Geert, De Pinte
  - Retie - PRAC De Vos, Axel, Dessel
  - Deurne - PRAC Heyvaert, Frank, Deurne
  - Deurne - PRAC Verelst, Joost, Deurne
  - Genk - PRAC Vernijns, J., Genk
  - Gozée - PRAC De Meulemeester, Marc, Gozée
  - Hasselt - PRAC Vantroyen, Daniel, Hasselt
  - Herent - PRAC Denolf, Bart, Herent
  - Linkebeek - PRAC Maury, Olivier, Linkebeek
  - Moorsel - PRAC Van Mulders, N., Moorsel
  - Natoye - PRAC Balthazar, Y., Natoye
  - Tremelo - PRAC Vermeersch, Lode, Tremelo
- Brazil (12):
  - Hospital Universitário João de Barros Barreto, Belém
  - Universidade Federal do Paraná, Curitiba
  - Hospital Geral de Goiânia Alberto Rassi, Goiânia
  - Centro de Pesquisas Clínicas Ltda, Higienópolis
  - Centro de Estudos em Diabetes e Hipertensão, Joaquim Távora
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Centro de Pesquisas em Diabetes, Porto Alegre
  - Instituto Estadual de Diabetes e Endocrinologia, Rio de Janeiro
  - Irmandade da Santa Casa de Misericórdia de São Paulo - IPEC - Instituto de Pesquisa Clínica, Santa Cecília
  - Instituto de Molestias Cardiovasculares - IMC, São José do Rio Preto
  - Hospital das Clinicas da FMUSP, São Paulo
  - Hospital do Rim e Hipertensão - UNIFESP, Vila Clementino
- Bulgaria (5):
  - Univ.Multiprofile Hospital "Dr. Georgy Stranski" EAD, Pleven, Pleven
  - Multiprofile Hospital for Active Treatment, Sofia
  - Multiprofile Hospital for Active Treatment "Zaritza Johanna", Sofia
  - Military Medical Academy, Clin. Endocrinology & Metab. Dis., Sofia
  - MHAT Prof Stoyan Kirkovich AD, Stara Zagora
- Canada (11):
  - IUCPQ (Laval University), Québec, Migration Data
  - First Line Medical Services Ltd., St. John's, Newfoundland and Labrador
  - Topsail Road Medical Clinic, St. John's, Newfoundland and Labrador
  - Cambridge Cardiac Care Inc., Cambridge, Ontario
  - Hamilton Medical Research Group, Hamilton, Ontario
  - SKDS Research Incorporated, Newmarket, Ontario
  - Wilderman Medical Clinic, Thornhill, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Albion Finch Medical Centre, Toronto, Ontario
  - Kings County Medical Centre, Montague, Prince Edward Island
  - Dynamik Research, Pointe-Claire, Quebec
- Chile (4):
  - Consulta Privada Maria Loreto Aguirre Coveña, Providencia
  - Hospital de Servicios Médicos Godoy Ltda, Providencia
  - Centro Medico Antulawen, Temuco
  - Hospital Naval Almirante Nef, Viña del Mar
- Colombia (11):
  - BioMelab, Barranquilla
  - Centro Cientifico Asistencial Jose Luis Accini, Barranquilla
  - Fundacion del Caribe de Investigacion Biomedica, Barranquilla
  - Dexa Diabetes Servicios Médicos Ltda, Bogotá
  - Endocare Research Institute, Bogotá
  - UNIENDO Unidad Integral de Endocrinologia, Bogotá
  - Centro cardiovascular Aristides, Cartagena
  - centro de Diagnostico Cardiologico para la Investigacion Bio, Cartagena
  - Fundacion Cardiovascular de Colombia, El Bosque
  - Fundación Oftalmologica de Santander, El Bosque
  - Fundación Centro de Investigaciones Biomédicas Riescard, Tolima
- Czechia (8):
  - Internal & Diabetology Ambulance, Jablonec nad Nisou, Jablonec nad Nisou
  - Diabetology & Internal Ambulance, Olomouc-Lazce
  - Internal & Diabetology Ambulance Dr. Vrkoc, Ostrava, Ostrava
  - Cardiology ambulance, Plzen, Pilsen
  - Diebetology internal Ambulance, Prague
  - ResTrial s.r.o., Prague
  - Internal & Diabetology Ambulance, Prostejov, Prostějov
  - Hospital Strakonice, Internal Department, Strakonice
- Finland (7):
  - Diabetesklinikka, Mehiläinen Töölö, Helsinki
  - Lääkärikeskus Ite, Joensuu
  - Lääkärikeskus Aava Kerava, Kerava
  - Kokkolan Lääkärikeskus, Kokkola
  - IteLasaretti, Kuopio
  - Terveystalo Oulu, Diapolis, Oulu
  - TYKS, Turku
- France (24):
  - CAB Hell M, MG, Behren Les Forbach, Behren-lès-Forbach
  - CAB Breton Dr Nicolas, Béziers
  - HOP Haut Levèque, Diabéto, Pessac, Bordeaux
  - CAB Lemarie B, MG, Bourg des Cptes, Bourg-des-Comptes
  - CAB Cadinot Dr D, Broglie, Broglie
  - CAB Ferrier R, MG, Cannes, Cannes
  - CAB Jordan E, MG, Carbonne, Carbonne
  - CAB Merlin P, MG Castets, Castets
  - CAB Fonteny R, MG, Chartres, Chartres
  - CAB Fournier P, MG, Chartres, Chartres
  - CAB Martocq G, MG, Cournonterral, Cournonterral
  - HOP, Fort de France, Fort de France, Fort de France
  - CAB Le Mouel S, MG, Hinx, Hinx
  - CAB Pholsena, MG, La Réunion, La Réunion
  - CAB Bismuth M, Labarthe-sur-Lèze
  - CAB Zimmermann D, Louvigne de Bie
  - CAB Mainetti P, MG, Maintenon, Maintenon
  - CAB Barucq F, MG, Orthez, Orthez
  - CAB Mostephai M, Orthez
  - CAB Cassagnes JL, MG, Palau Del Vidre, Palau-del-Vidre
  - CAB Mercey Y, MG, St Genies des Fontaines, Saint Genies Des Fontaines
  - Hop St Dié des Vosges, Diabéto, St Dié des Vosges, Saint-Dié
  - CAB Bonneau D, MG, Thouars, Thouars
  - CAB Morel H, MG, Tilly sur Seulles, Tilly-sur-Seulles
- Georgia (10):
  - Unimed Ajara LLC, Private Practice, Batumi
  - Central Hospital LTD 'Gormedi', Gori, Gori
  - L&J Clinic, Kutaisi, Kutaisi
  - EC Cardiology Clinic,Tbilisi, Tbilisi
  - National Center for Diabetes Research Ltd., Tbilisi, Tbilisi
  - National Institute of Endocrinology, Tbilisi, Tbilisi
  - Zhordania Institute of Human Reproduction, Tbilisi, Tbilisi
  - Medical Centre Medelite Ltd., Tbilisi, Tbilisi
  - Chemotherapy & Immunotherapy Clinic 'Medulla', Tbilisi, Tbilisi
  - JSC 'Curatio', Zugdidi
- Germany (39):
  - Universitätsklinikum Aachen, AöR, Aachen
  - Studienzentrum Klausmann, Aschaffenburg
  - Gemeinschaftspraxis, Asslar, Aßlar
  - Diabetes Schwerpunktpraxis, Bad Nauheim
  - Praxis Dr. Naumburger, Berlin, Berlin
  - emovis GmbH, Berlin
  - Praxis Dr. Rieker, Berlin, Berlin
  - IFG Institut für Gesundheitsförderung GmbH, Berlin
  - Dünnwaldpraxis, Köln, Cologne
  - MVZ DaVita Dormagen GmbH, Dormagen- Hackenbroich
  - Praxis Dr. Busch, Dortmund, Dortmund
  - GWT-TUD GmbH, Dresden
  - Praxis Dr. Schlecht, Eisenach, Eisenach
  - ZKS Südbrandenburg GmbH, Elsterwerda
  - Praxis Dr. Huptas, Essen, Essen
  - Praxis Dr. Schmidt, Flörsheim, Flörsheim
  - Institut für Stoffwechselforschung, Frankfurt, Frankfurt
  - Praxis Dr. Groeneveld, Furth im Wald, Furth im Wald
  - Praxis Dr. Kohlhas, Gebhardshain, Gebhardshain
  - Praxis Dr. Samer, Haag, Haag
  - Klinische Forschung Management & Services GmbH, Hamburg
  - Diabetologische Schwerpunktpraxis, Hamburg
  - Praxis Dr. Burkhardt, Hamburg, Hamburg
  - Diabeteszentrum Alstertal, Hamburg, Hamburg
  - Praxis Dr. Herrmann, Hatten, Kirchhatten
  - Praxis Dr. Klein, Künzing, Künzing
  - Praxis Dr. Nischik, Leipzig, Leipzig
  - Praxis Dr. Kropp, Lübeck, Lübeck
  - PFÜTZNER Science & Health Institute GmbH, Mainz
  - Diabetologische Schwerpunktpraxis, Münster
  - Praxis Dr. Böckmann, Neumünster
  - Praxis Dr. Hilgenberg, Rehburg-Loccum
  - Praxis Dr. Naudts, Rodgau, Rodgau/Dudenhofen
  - Praxis Dr. Hirschhäuser, Saarbrücken
  - Praxis Dr. Segner, St. Ingberg, Saint Ingbert / Oberwürzbach
  - Praxis Dr. Herrmann, Schwabenheim
  - Praxis Dr. Dietlein, Stadtbergen
  - Praxis Dr. Sauter, Wangen
  - Schwerpunktpraxis Diabetologie, Zwenkau
- Greece (8):
  - General Hospital of Athens Evangelismos, Athens
  - General University Hospital "Attikon", Haidari, Athens
  - Univ. Gen. Hosp. of Ioannina, Ioannina
  - General Hospital "Amalia Fleming", Melissia, Athens
  - General Hospital of Nikaia, Nikaia
  - University General Hospital of Thessaloniki AHEPA, Thessaloniki
  - General Hopsital of Thessaloniki "Ippokrateio", Thessaloniki
  - Kliniki Thermi, Thessaloniki
- Hong Kong (3):
  - Alice Ho Miu Ling Nethersole Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Hungary (9):
  - Imre Magyar Hospital, Ajka, Ajka
  - Lausmed Kft. Outpatient Unit of Internal Medicine, Baja
  - Karolyi Sandor Hospital, Budapest, Budapest
  - Bekes County Pandy Kalman Hospital, Gyula
  - Erzsebet Hospital, Hodmezövasarhely, Hódmezövásárhely
  - Dr. Samuel Diosszilagyi Hospital and Outpatient Clinic, Mako, Makó
  - TaNa Med Kft., Mosonmagyaróvár
  - Grof Esterhazy Hospital and Outpatient Clinic, Pápa
  - Tolna County Balassa Janos Hospital, Szekszárd
- India (24):
  - Shree Krishna Hospital and Heart Care Centre, Ahmedabad, Ahmedabad
  - CIIGMA Institute of Medical Sciences Pvt Ltd, Aurangabad
  - Diabetes care and research centre, Bangalore
  - Manipal Hospital, Bangalore
  - Bangalore Diabetes Centre (BDC)- Medisys Clinical Research, Bangalore
  - MS Ramaiah Memorial Hospital,, Bangalore, Karnataka
  - Belgaum Diabetes Centre, Belgaum, Belagavi
  - Swamy Diabetes Centre, Chennai
  - Apollo Hospitals, Chennai
  - M V Hospital For Diabetes and Diabetes Research Centre, Chennai
  - Dr. Mohans Diabetes Speciality Centre, Chennai
  - Kovai Diabetes Speciality Centre & Hospital, Coimbatore
  - TOTALL Diabetes Hormone Institute, Indore
  - Diabetes Thyroid and Endocrine Centre, Jaipur
  - Diamed Clinical Research Services Pvt. Ltd., Jaipur
  - Grant Medical Foundation, Ruby Hall Clinic, Maharashtra
  - Global Hospital- Superspeciality & Transplant Centre, Mumbai
  - RHIDEM, Mumbai
  - K.G.N. Diabetes and Endocrine Centre, Mumbai, Maharastra
  - Sunil's Diabetes care and Research Centre, Nagpur
  - Jahingir Clinical Development Centre, Pune
  - Deshmukh Clinic, Pune
  - Diabetes Care Center, Thiruvananthapuram
  - Yalamanchi Hospitals & Research Centres Pvt Ltd., Vijayawada
- Ireland (4):
  - The Red House Family Practice, Co. Cork
  - Connolly Hospital Blanchardstown, Dublin
  - The Palms GP Surgery, Gorey
  - Fethard-on-Sea Medical Practice, Wexford
- Israel (7):
  - Barzilai Medical Center, Ashkelon
  - Rambam Medical Center, Haifa
  - Edith Wolfson Medical Center, Diabetic Unit, Holon, Holon
  - Hadassah Medical Center, Ein-Karem, Jerusalem
  - Western Galilee Hospital, Nahariya
  - Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center Tel Hashomer, Tel Litwinsky
- Italy (9):
  - Ospedale "SS. Trinità", Cagliari
  - Policlinico Universitario Mater Domini, Universita di Catanzaro, Catanzaro
  - Policlinico San Martino, Genova
  - Ospedale di Guastalla, Guastalla (RE)
  - A.O.U.Policlinico G.Martino, Messina
  - Fondazione Centro San Raffaele del Monte Tabor, Milan
  - Ospedale S. Pertini, Roma
  - Azienda Ospedaliera Sant'Andrea-Università di Roma La Sapienza, Roma
  - IRCCS Gruppo Multimedica, Sesto San Giovanni (MI)
- Japan (14):
  - Daishinkai Medical Corporation Ookuma Hospital, Aichi, Nagoya
  - Chibanishi General Hospital, Chiba, Matsudo
  - New Tokyo Heart Clinic, Chiba, Matsudo
  - Kashinoki I.M. Clinic, Fukushima, I.M., Fukushima, Date
  - Japan Community Health care Organization Nihonmatsu Hospital, Fukushima, Nihonmatsu
  - Iwase General Hospital, Fukushima, Sukagawa
  - Iryohojinshadan Sasaki Clinic, Hyogo, Amagasaki
  - Takasagoseibu Hospital, Hyogo, Takasago
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa, Yokohama
  - Jinnouchi Clinic Diabetes Care Center, Kumamoto, Kumamoto
  - Kumamoto Rosai Hospital, Kumamoto, Yatsushiro
  - Koga General Hospital, Miyazaki, Miyazaki
  - Saitama Medical Cooperative Association Hanyu General Hospital, Saitama, Hanyu
  - Nihon University Itabashi Hospital, Tokyo, Itabashi-ku
- Malaysia (8):
  - Penang Medical College, George Town
  - Monash University, Johor Bahru, Johor
  - Hospital University Sains Malaysia, Kota Bharu
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Hospital Melaka, Malacca
  - Hospital Taiping, Taiping
- Mexico (5):
  - Hospital General de Acapulco, Acapulco
  - Centro de Investigacion Cardiometabolica de Aguascalientes, Aguascalientes
  - Instituto Nacional de Cardiologia Ignacio Chavez, Distrito Federal
  - Unidad de Investigacion Clinica Cardiometabolica de Occident, Guadalajara
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
- Netherlands (16):
  - Huisartspraktijk Emmers, 's-Hertogenbosch
  - FlevoResearch, Almere Stad
  - Academisch Medisch Centrum (AMC), Amsterdam
  - Rode Kruis Ziekenhuis Beverwijk, Beverwijk
  - Andromed Breda, Breda
  - Noordwest Ziekenhuisgroep, location Den Helder, Den Helder
  - Andromed Eindhoven, Eindhoven
  - Andromed Noord, Groningen
  - Vasculair Onderzoek Centrum, Hoorn
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Andromed Rotterdam, Rotterdam
  - Rotterdam Research Institute, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
  - Antonius Ziekenhuis, Sneek
  - Andromed Oost, Velp
  - Andromed Leiden-Zoetermeer, Zoetermeer
- New Zealand (4):
  - Christchurch Hospital, Christchurch
  - RMC Medical Research Ltd, Dunedin
  - P3 Research, Wellington, Newtown Wellington NZ
  - P3 Research, Promed House, Tauranga
- Norway (11):
  - Medi 3 AS, Ålesund
  - Bodø Legesenter AS, avd. for med. studier, Bodø
  - Medi 3 Innlandet AS, avd Elverum, Elverum
  - Vestre Viken HF, Bærum sykehus, Gjettum
  - M3 Helse AS, Hamar
  - Bylegene SA, Jessheim
  - Heiaklinikken, Lierskogen
  - Rådhuset Spesialistsenter, Oslo
  - Sandvika Spesialistsenter, Sandvika
  - Grålum Legesenter, Sarpsborg
  - Forusakutten - Kolibri Medical, Avd. Stavanger, Stavanger
- Peru (8):
  - Instituto Delgado de Investigacion Medica, Arequipa
  - Clinica San Pedro, Huacho
  - Hospital Nacional Dos de Mayo, Lima
  - Clinica Internacional, Lima
  - Centro de Investigaciones Médicas METABOLICARE SAC, Lima
  - Clinica San Gabriel, Lima
  - Centro De Especialidades Medicas Santa Maria S.A.C, Piura
  - Clinica San Judas Tadeo, San Miguel
- Philippines (10):
  - Asian Hospital & Medical Center, City of Muntinlupa
  - Center for Diabetes Care, Iloilo City
  - Mary Mediatrix Medical Center, Lipa City, Batangas
  - Philippine General Hospital, Manila
  - University of Santo Tomas Hospital, Manila
  - Manila Doctors Hospital, Manila
  - St. Luke's Medical Center, Quezon City
  - Quirino Memorial Medical Center, Quezon City
  - Cardinal Santos Medical Center, San Juan City
  - Surigao Health Specialists, Surigao City
- Portugal (8):
  - Hospital Fernando Fonseca, EPE, Amadora
  - CHLO, EPE - Hospital de Santa Cruz, Carnaxide
  - CHUC - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - Centro Hospitalar da Cova da Beira Hospital Pêro da Covilhã, Covilha
  - Hospital Distrital Figueira da Foz, EPE, Figueira da Foz Municipality
  - Hospital da Luz, Lisbon
  - Centro Hospitalar São João,EPE, Porto
  - Centro Hospitalar de Entre o Douro e Vouga, E.P.E. - Hospital de São Sebastião, Santa Maria da Feira
- Romania (6):
  - SC Diabol SRL, Brasov, Brasov
  - Nicodiab SRL, Bucharest, Bucharest
  - SC Medical Centre "Sanatatea Ta" SRL, Bucharest, Bucharest
  - Consultmed SRL, Iasi, Iași
  - Emergency County Clinical Hospital, Sibiu, Sibiu
  - Private Practice Dr. Remus Gagiu, Târgovişte
- Russia (9):
  - LLC Clinic of new technologies of medicine, Dzerzhinsky
  - City Clinical Hospital No. 6 of MoH of Udmurt Republic, Izhevsk
  - City Clinical Hospital No. 4, Moscow, Moscow
  - City Clinical Hospital No. 13, Moscow, Moscow
  - State Institution "Central Clinical Hospital of RAS", Moscow, Moscow
  - City Clinical Hospital No. 61, Moscow, Moscow
  - State Healthcare Institution, Regional hospital #2, Rostov-on-Don
  - Limited Liability Company "CENTER DIABET", Samara, Samara
  - MMU City Outpatient Clinic no. 20, Saratov, Saratov
- Serbia (5):
  - Clinical Medical Center Zvezdara, Belgrade, Belgrade
  - Clinical Centre Nis, Niš
  - General Hospital Pancevo, Pančevo
  - General Hospital Subotica, Internal Medicine, Subotica
  - Clinical Hospital Center Zemun, Zemun
- Slovakia (7):
  - DIASTYLE s.r.o., Diabetology Outpatient Department, Banská Bystrica
  - ENDIAMED s.r.o., Dolny Kubin, Dolný Kubín
  - CELL B s.r.o., Levice
  - DIA-KONTROL s.r.o., Levice
  - Funkystuff s.r.o., Nove Zamky, Nové Zámky
  - Diabetologicka ambulancia MUDr. Lucia Gajdosikova s.r.o., Považská Bystrica
  - MEDIVASA s.r.o., Outpatient Clinic, Zilina, Žilina
- South Africa (10):
  - Dr. P. Patel, Cape Town
  - Dr. E. L. Janari, Cape Town
  - Dr. Vawda, Durban
  - Parklands Medical Centre, Durban
  - Dr. Jurgens, Krugersdorp
  - Dr. H. Makan, Lenasia
  - Dr. D. R. Lakha, Johannesburg, Lenasia
  - Greenacres Hospital, Port Elizabeth
  - Dr. M. Seeber, Pretoria
  - Vergelegen Medi-Clinic, Somerset West
- South Korea (15):
  - Korea University Ansan Hospital, Ansan
  - Inje University Busan Paik Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - National Health Insurance Service Ilsan Hospital, Goyang
  - Dongguk University Ilsan Hospital, Goyang
  - Inje University Ilsan Paik Hospital, Goyang
  - Chonbuk National University Hospital, Jeonju
  - Pusan National Univ. Hosp, Pusan
  - Seoul National University Bundang Hospital, Seongnam
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Wonju Severance Christian Hosp, Wŏnju
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (18):
  - C.A.P. Sardenya, Barcelona
  - CAP Les Corts, Barcelona
  - CAP Casanova, Barcelona
  - CAP Burjassot 1, Burjassot
  - C.S. Natahoyo, Gijón
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - CAP Florida, L'Hospitalet de Llobregat
  - Hospital de Bellvitge, L'Hospitalet de Llobregat
  - CAP La Roca, La Roca Del Vallés (Barcelona)
  - Hospital General Universitario Gregorio Marañón, Madrid
  - C.S. El Cristo, Oviedo
  - C.S. Colloto, Oviedo
  - C.S. Vallobin-La Florida, Oviedo
  - ABS Pineda de Mar, Pineda de Mar
  - Hospital de l'Esperit Sant, Santa Coloma de Gramanet
  - CAP Tàrrega, Tàrrega
  - CS Ingeniero Joaquin Benlloch, Valencia
  - Hospital Clínico de Valencia, Valencia
- Sweden (9):
  - CTC Sahlgrenska Universitetssjukhuset, Gothenburg
  - Sjukhuset, Härnösand, Härnösand
  - Avonova Hälsa AB, Järfälla
  - Skånes universitetssjukhus, Malmö, Malmo
  - Dalecarlia Clinical Research Center, Rättvik
  - Södra Dalarnas vårdcentral, Hedemora, Rättvik
  - Näsets Läkargrupp, Skanör
  - Vårdcentralen Silentzvägen, Uddevalla
  - S3 Clinical Research Centers, Vällingby
- Switzerland (4):
  - Allgemeine Medizin, Basel
  - FMH endocrinologia diabetologia, Bellinzona
  - Inselspital Bern, Bern
  - Dr. Pietro Gerber, Lugano
- Taiwan (15):
  - Chang-Hua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - E-Da Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - NCKUH, Tainan
  - National Taiwan University Hospital, Taipei
  - Shih-Kong Wu Ho-Shu Memorial Hospital, Taipei
  - Taipe Veterans General Hospital, Taipei
  - Cheng Hsin General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Cardinal Tien Hospital, Taipei
  - Taipei Medical University-Shuang Ho Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
- Tunisia (4):
  - HOP Fattouma Bourguiba, Mint, Monastir, Monastir
  - HOP Hédi Chaker, Endo, Sfax, Sfax
  - HOP Farhat Hached, Mint, Sousse, Sousse
  - HOP Habib Thameur, Mint, Tunis, Tunis
- Ukraine (10):
  - Donetsk Regional Clinical Hosp, Therapy Department, Donetsk
  - Ivano-Frankivsk City Central Clinical Hospital, Ivano-Frankivsk
  - City Clinical Hospital No. 27, Kharkiv, Kharkiv
  - City Clinical Hospital No. 17, Kharkov, Kharkiv
  - Clinic for Cardiology "Sertse i sudyny", Kiev, Kiev
  - City Clinical Hospital No. 1, Kiev, Kiev
  - Poliklinika #2, Kyiv, Kyiv
  - City Hospital No. 5, Lvov, Lviv
  - Odeska zaliznichna likarnya, Odessa, Odesa
  - Vinnitsia Regional Endocrinology Dispensary, Vinnitsa
- United Kingdom (10):
  - Crouch Oak Family Practice, Addlestone
  - Ash Vale Health Centre, Aldershot, Ash Vale, Aldershot
  - Birmingham Heartlands Hospital, Birmingham
  - Hathaway Medical Centre, Chippenham
  - University Hospital of North Durham, Durham
  - St Mary's Surgery, Ely
  - Gloucestershire Royal Hospital, Gloucester
  - James Paget University Hospital, Great Yarmouth
  - Morriston Hospital, Swansea
  - Royal Cornwall Hospital, Truro

REFERENCES:
- [Derived] Marx N, Kolkailah AA, Rosenstock J, Johansen OE, Cooper ME, Alexander JH, Toto RD, Wanner C, Espeland MA, Mattheus M, Schnaidt S, Perkovic V, Gollop ND, McGuire DK. Hypoglycemia and Cardiovascular Outcomes in the CARMELINA and CAROLINA Trials of Linagliptin: A Secondary Analysis of Randomized Clinical Trials. JAMA Cardiol. 2024 Feb 1;9(2):134-143. doi: 10.1001/jamacardio.2023.4602. PMID 38170502
- [Derived] Balasubramanian P, Kernan WN, Sheth KN, Ofstad AP, Rosenstock J, Wanner C, Zinman B, Mattheus M, Marx N, Inzucchi SE. Baseline Cardiovascular Risk Factor Control in Patients With Type 2 Diabetes and Coronary Disease Versus Stroke: Secondary Analysis of Cardiovascular Outcome Trials. Stroke. 2023 Aug;54(8):2013-2021. doi: 10.1161/STROKEAHA.122.042053. Epub 2023 Jul 14. PMID 37449424
- [Derived] Dar MS, Wanner C, Marx N, Ofstad AP, Mattheus M, Kaspers S, Beg SA. Cardiovascular outcomes trial data from EMPA-REG OUTCOME, CAROLINA and CARMELINA: Assessment of a novel staging system for type 2 diabetes. Diabetes Obes Metab. 2023 May;25(5):1372-1384. doi: 10.1111/dom.14989. Epub 2023 Mar 6. PMID 36700391
- [Derived] Verhagen C, Janssen J, Minderhoud CA, van den Berg E, Wanner C, Passera A, Johansen OE, Biessels GJ. Chronic kidney disease and cognitive decline in patients with type 2 diabetes at elevated cardiovascular risk. J Diabetes Complications. 2022 Oct;36(10):108303. doi: 10.1016/j.jdiacomp.2022.108303. Epub 2022 Aug 31. PMID 36116359
- [Derived] Verhagen C, Janssen J, Biessels GJ, Johansen OE, Exalto LG. Females with type 2 diabetes are at higher risk for accelerated cognitive decline than males: CAROLINA-COGNITION study. Nutr Metab Cardiovasc Dis. 2022 Feb;32(2):355-364. doi: 10.1016/j.numecd.2021.10.013. Epub 2021 Oct 27. PMID 34895804
- [Derived] Biessels GJ, Verhagen C, Janssen J, van den Berg E, Wallenstein G, Zinman B, Espeland MA, Johansen OE. Effects of linagliptin vs glimepiride on cognitive performance in type 2 diabetes: results of the randomised double-blind, active-controlled CAROLINA-COGNITION study. Diabetologia. 2021 Jun;64(6):1235-1245. doi: 10.1007/s00125-021-05393-8. Epub 2021 Feb 9. PMID 33559704
- [Derived] Rosenstock J, Kahn SE, Johansen OE, Zinman B, Espeland MA, Woerle HJ, Pfarr E, Keller A, Mattheus M, Baanstra D, Meinicke T, George JT, von Eynatten M, McGuire DK, Marx N; CAROLINA Investigators. Effect of Linagliptin vs Glimepiride on Major Adverse Cardiovascular Outcomes in Patients With Type 2 Diabetes: The CAROLINA Randomized Clinical Trial. JAMA. 2019 Sep 24;322(12):1155-1166. doi: 10.1001/jama.2019.13772. PMID 31536101
- [Derived] Janssen J, van den Berg E, Zinman B, Espeland MA, Geijselaers SLC, Mattheus M, Johansen OE, Biessels GJ. HbA1c, Insulin Resistance, and beta-Cell Function in Relation to Cognitive Function in Type 2 Diabetes: The CAROLINA Cognition Substudy. Diabetes Care. 2019 Jan;42(1):e1-e3. doi: 10.2337/DC18-0914. No abstract available. PMID 30811335
- [Derived] Chilton R. Linagliptin versus glimepiride add-on for the long-term treatment of Type 2 diabetes mellitus. Expert Rev Endocrinol Metab. 2013 Jul;8(4):345-349. doi: 10.1586/17446651.2013.811849. PMID 30736150
- [Derived] Biessels GJ, Janssen J, van den Berg E, Zinman B, Espeland MA, Mattheus M, Johansen OE; CAROLINA(R) investigators. Rationale and design of the CAROLINA(R) - cognition substudy: a randomised controlled trial on cognitive outcomes of linagliptin versus glimepiride in patients with type 2 diabetes mellitus. BMC Neurol. 2018 Jan 15;18(1):7. doi: 10.1186/s12883-018-1014-7. PMID 29334906
- [Derived] Marx N, Rosenstock J, Kahn SE, Zinman B, Kastelein JJ, Lachin JM, Espeland MA, Bluhmki E, Mattheus M, Ryckaert B, Patel S, Johansen OE, Woerle HJ. Design and baseline characteristics of the CARdiovascular Outcome Trial of LINAgliptin Versus Glimepiride in Type 2 Diabetes (CAROLINA(R)). Diab Vasc Dis Res. 2015 May;12(3):164-74. doi: 10.1177/1479164115570301. Epub 2015 Mar 15. PMID 25780262

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicentre, multinational, randomised, double-blind, double-dummy, parallel group,comparator-controlled trial compared Linagliptin versus (vs.) Glimepiride, predominantly on metformin background treatment in participants with type 2 diabetes mellitus (T2DM) at elevated cardiovascular (CV) risk receiving usual care.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended specialist sites which would then ensure that all participants met all inclusion/exclusion criteria. Participants were not to be randomised to trial treatment if any one of the specific entry criteria were not met.
Groups:
- Linagliptin: After 2-4 weeks placebo run-in phase, participants were administered 1 tablet of 5 milligram (mg) linagliptin plus 1 over-encapsulated tablet of placebo matching glimepiride, which was uptitrated in 4-week intervals during the first 16 weeks of treatment to the next dose. Both doses were administered once daily orally up to an estimated 432 weeks treatment period.
- Glimepiride: After 2-4 weeks placebo run-in phase, participants were administered 1 tablet of placebo matching linagliptin plus 1 over-encapsulated tablet of 1 to 4 mg glimepiride, which was uptitrated in 4-week intervals during the first 16 weeks of treatment to the next dose. Both doses were administered once daily orally up to an estimated 432 weeks treatment period.
Period: Discontinuation From Study (Treated Set)
Arm/Group | Linagliptin | Glimepiride
Started (Started are entered/ randomised) | 3028 | 3014
Patient Died (Other Cause Than CV Death) | 123 | 146
Treated | 3023 | 3010
Completed (Completed regarding MACE status or died) | 2899 | 2895
Not Completed | 129 | 119
Not completed — Consent Withdrawn (Status Alive) | 49 | 37
Not completed — Consent Withdrawn (Status Unknown) | 14 | 12
Not completed — Site Closure (Status Alive) | 15 | 22
Not completed — Site Closure (Status Unknown) | 0 | 1
Not completed — LostToFollowUpfor3P-MACE(StatusAlive) | 38 | 35
Not completed — LostToFollowUpfor3P-MACE(StatusUnknown) | 8 | 8
Not completed — Not treated | 5 | 4
Period: Discontinuation From Treatment
Arm/Group | Linagliptin | Glimepiride
Started (Started are entered/ randomised) | 3028 | 3014
Treated | 3023 | 3010
Completed (Not prematurely discontinued from trial medication) | 1896 | 1832
Not Completed | 1132 | 1182
Not completed — Not treated | 5 | 4
Not completed — Adverse Event | 457 | 523
Not completed — Lack of Efficacy | 61 | 41
Not completed — Protocol Violation | 46 | 47
Not completed — Lost to Follow-up | 24 | 28
Not completed — Withdrawal by Subject | 309 | 328
Not completed — Other than listed above | 230 | 211

BASELINE CHARACTERISTICS:
Population: Treated set (TS): All patients treated with at least one dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Linagliptin | Glimepiride | Total
Number analyzed (Participants) | 3023 | 3010 | 6033
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (9.5) | 64.2 (9.5) | 64.0 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1185 | 1229 | 2414
  Male | 1838 | 1781 | 3619
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 519 | 513 | 1032
  Not Hispanic or Latino | 2495 | 2487 | 4982
  Unknown or Not Reported | 9 | 10 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 106 | 108 | 214
  Asian | 531 | 530 | 1061
  Native Hawaiian or Other Pacific Islander | 5 | 3 | 8
  Black or African American | 155 | 169 | 324
  White | 2217 | 2190 | 4407
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: The First 3-point Major Adverse Cardiovascular Events (3P-MACE)
Description: The first occurrence of any of the following Clinical Event Committee (CEC) confirmed adjudicated components of the primary composite endpoint: CV death (including fatal stroke and fatal myocardial infarction (MI)), non-fatal MI (excluding silent MI), or nonfatal stroke is presented.
Time Frame: From randomization until individual day of trial completion, up to 432 weeks
Population: Treated set (TS): All patients treated with at least one dose of trial drug.
Measure: Number; unit: Events/ 1000 patients-years
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 3023 | 3010
Events/ 1000 patients-years | 20.7 | 21.2
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; Test type: Non-Inferiority — This was the first step in a pre-defined hierarchical testing approach. The upper bound of the confidence interval (CI) of the Hazard ratio (HR) of linagliptin vs. glimepiride was compared with this noninferiority margin for the testing of non-inferiority. All non-inferiority tests were based on a margin of 1.3; p < 0.0001, Regression, Cox — P-values derived from Wald´s Chi-square test for non-inferiority were calculated; Cox proportional-hazard model with factor treatment was applied to compare linagliptin with glimepiride; Hazard Ratio (HR) = 0.98, 95.47% CI 2-sided [0.84 to 1.14]
Statistical Analysis 2: Comparison: Linagliptin vs Glimepiride; Test type: Superiority — This was the second step in a pre-defined hierarchical testing approach; p = 0.3813, Regression, Cox — P-values derived from Wald´s Chi-square test; Cox proportional-hazard model with factor treatment was applied to compare linagliptin with glimepiride; Hazard Ratio (HR) = 0.98, 95.47% CI 2-sided [0.84 to 1.14]

2. Secondary Outcome: The First 4-point (4P)- MACE
Description: The first key secondary endpoint was time to first occurrence of any of the following adjudicated components of the composite endpoint: CV death (including fatal stroke and fatal MI), non-fatal stroke, non-fatal MI (excluding silent MI), or hospitalisation for unstable angina pectoris.
Time Frame: From randomization until individual day of trial completion, up to 432 weeks
Population: TS
Measure: Number; unit: Events/ 1000 patients-years
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 3023 | 3010
Events/ 1000 patients-years | 23.4 | 23.7
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; Test type: Superiority — This was the third step in a pre-defined hierarchical testing approach; p = 0.4334, Regression, Cox — P-values derived from Wald´s Chi-square test for non-inferiority; Cox proportional-hazard model with factor treatment was applied to compare linagliptin with glimepiride; Hazard Ratio (HR) = 0.99, 95.47% CI 2-sided [0.86 to 1.14]

3. Secondary Outcome: Percentage of Participants Taking Trial Medication at Trial End, Maintained Glycaemic Control (HbA1c ≤7.0%) Without Need for Rescue Medication, Without >2% Weight Gain, and Without Moderate/Severe Hypoglycaemic Episodes During Maintenance Phase
Description: The second key secondary endpoint was a composite endpoint of treatment sustainability, defined as the percentage of patients taking trial medication at trial end, maintained glycaemic control (HbA1c ≤7.0%) without need for rescue medication, without >2% weight gain, and without moderate/severe hypoglycaemic episodes during maintenance phase.
Time Frame: From Visit 6 (Week 16) to Final visit (Week 432) (Maintenance Phase)
Population: TS without duplicates (TS w/o duplicates), patients who are off-drug or died prior to regular study stop were handled as non-completers considered failure (NCF).
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 3014 | 3000
Percentage of participants (%) | 16.0 [14.7 to 17.3] | 10.2 [9.1 to 11.3]
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; Test type: Other; p < 0.0001, Regression, Logistic — p-value derived from logistic regression; Odds Ratio (OR) = 1.68, 95.47% CI 2-sided [1.43 to 1.96] — Odds ratio and confidence interval are based on logistic regression with factor for treatment

4. Secondary Outcome: Percentage of Participants Who Were on Trial Medication at Trial End, Maintained Glycaemic Control (HbA1c ≤7.0%) Without Need for Rescue Medication, and Without >2% Weight Gain During Maintenance Phase
Description: The third key secondary endpoint was a composite endpoint of treatment sustainability, defined as percentage of patients who were on trial medication at trial end, maintained glycaemic control (HbA1c ≤7.0%) without need for rescue medication, and without >2% weight gain during maintenance phase.
Time Frame: From Visit 6 (Week 16) to Final visit (Week 432) (Maintenance Phase)
Population: TS w/o duplicates (NCF)
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 3014 | 3000
Percentage of participants (%) | 17.4 [16.1 to 18.8] | 14.1 [12.9 to 15.4]
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; This was the fifth step in a pre-defined hierarchical testing approach; Test type: Other; p = 0.0004, Regression, Logistic — p-value derived from logistic regression; Odds Ratio (OR) = 1.29, 95.47% CI 2-sided [1.11 to 1.48] — Odds ratio and confidence interval are based on logistic regression with factor for treatment

5. Secondary Outcome: Percentage of Participants With the Occurrence of at Least One Event of 3P-MACE
Description: Percentage of participants occurrence of at least one of the following adjudicated components of CV death (including fatal stroke and fatal MI), non-fatal MI (excluding silent MI) and non-fatal stroke is presented as secondary CV endpoint.
Time Frame: From randomization until individual day of trial completion, up to 432 weeks
Population: TS
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 3023 | 3010
Percentage of participants (%) | 11.8 [10.7 to 13.0] | 12.0 [10.9 to 13.2]

6. Secondary Outcome: Percentage of Participants With the Occurrence of at Least One Event of 4P -MACE
Description: Percentage of participants occurrence of at least one of the following adjudicated components of CV death (including fatal stroke and fatal MI), non-fatal MI (excluding silent MI), non-fatal stroke, and hospitalisation for unstable angina pectoris is presented as secondary CV endpoint.
Time Frame: From randomization until individual day of trial completion, up to 432 weeks
Population: TS
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 3023 | 3010
Percentage of participants (%) | 13.2 [12.0 to 14.4] | 13.3 [12.2 to 14.6]

7. Secondary Outcome: Percentage of Participants With Occurrence of Any of the Components of the Composite Endpoint of All Adjudication-confirmed Events
Description: Percentage of participants with occurrence of any of the following components of the composite endpoint of all adjudication-confirmed events of:
  * CV death (including fatal stroke and fatal MI)
  * non-fatal MI
  * non-fatal stroke
  * hospitalisation for unstable angina pectoris
  * TIA
  * hospitalisation for heart failure
  * hospitalisation for coronary revascularisation procedures (CABG, PCI)
Time Frame: From start of the treatment until 7 days after the end of treatment, up to 433 weeks
Population: TS
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 3023 | 3010
Percentage of participants (%) | 17.1 [15.8 to 18.5] | 17.8 [16.4 to 19.2]

8. Secondary Outcome: Time to First Occurrence of Any of the Components of the Composite Endpoint of All Adjudication-confirmed Events
Description: Time to first occurrence of any of the following components of the composite endpoint of all adjudication-confirmed events of:
  * CV death (including fatal stroke and fatal MI)
  * non-fatal MI
  * non-fatal stroke
  * hospitalisation for unstable angina pectoris
  * Transient ischaemic attack (TIA)
  * hospitalisation for heart failure
  * hospitalisation for coronary revascularisation procedures (CABG, PCI)
Time Frame: From start of the treatment until 7 days after the end of treatment, up to 433 weeks
Population: TS
Measure: Number; unit: Events/ 1000 patients-years
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 3023 | 3010
Events/ 1000 patients-years | 31.1 | 32.4
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; This was the fifth step in a pre-defined hierarchical testing approach; Test type: Other; p = 0.5249, Regression, Cox — p-value derived from Wald´s chi-square test; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.85 to 1.09] — Hazard ratio and confidence interval derived from Cox regression with factor treatment

9. Secondary Outcome: Change From Baseline to Final Visit in Hemoglobin A1c (HbA1c)
Description: Change from baseline to final visit in HbA1c is presented as secondary diabetes-related endpoint. Least square mean is adjusted mean. The Final Visit value referred to the last value obtained on-treatment.
Time Frame: Baseline and week 432
Population: TS w/o duplicates considering all available data
Measure: Least Squares Mean (Standard Error); unit: Percentage glycosylated hemoglobin (%)
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 2951 | 2949
Percentage glycosylated hemoglobin (%) | 0.06 (0.02) | 0.15 (0.02)
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; This was the fifth step in a pre-defined hierarchical testing approach; Test type: Other; p = 0.0023, ANCOVA; The Analysis of Covariance (ANCOVA) model includes the fixed categorical effect of treatment and the continuous covariate of baseline HbA1c; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.15 to -0.03], Standard Error of Mean 0.03 — Mean difference = Linagliptin mean - Glimepiride mean

10. Secondary Outcome: Change From Baseline to Final Visit in Fasting Plasma Glucose (FPG)
Description: Change from baseline to final visit in fasting plasma glucose (FPG) is presented as secondary diabetes-related endpoint. Least square mean is adjusted mean. The Final Visit value referred to the last value obtained on-treatment.
Time Frame: Baseline and week 432
Population: TS w/o duplicates considering all available data
Measure: Least Squares Mean (Standard Error); unit: Milligram/ deciliter (mg/dL)
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 2996 | 2949
Milligram/ deciliter (mg/dL) | 12.4 (0.9) | 19.7 (0.9)
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; This was the fifth step in a pre-defined hierarchical testing approach; Test type: Other; p < 0.0001, ANCOVA; The ANCOVA model includes the fixed categorical effect of treatment and the continuous covariate of baseline FPG; Mean Difference (Final Values) = -7.3, 95% CI 2-sided [-9.7 to -4.8], Standard Error of Mean 1.2 — Mean difference = Linagliptin mean - Glimepiride mean

11. Secondary Outcome: Change From Baseline to Final Visit Fasting Total Cholesterol, Low-density Lipoprotein (LDL) Cholesterol and High-density Lipoprotein (HDL) Cholesterol
Description: Change from baseline to final visit in total cholesterol, low-density lipoprotein (LDL) cholesterol and high-density lipoprotein (HDL) cholesterol is presented as secondary diabetes-related endpoint. Least square mean is adjusted mean. The Final Visit value referred to the last value obtained on-treatment.
Time Frame: Baseline and week 432
Population: TS w/o duplicates, participants on treatment
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 3014 | 3000
mg/dL
  LDL cholesterol: number analyzed (Participants) | 2688 | 2660
  LDL cholesterol | -6.1 (0.6) | -6.5 (0.6)
  HDL cholesterol: number analyzed (Participants) | 2783 | 2751
  HDL cholesterol | 0.7 (0.2) | 0.3 (0.2)
  Total cholesterol: number analyzed (Participants) | 2788 | 2762
  Total cholesterol | -5.4 (0.7) | -0.5 (0.7)
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; LDL cholesterol, this was the fifth step in a pre-defined hierarchical testing approach; Test type: Other; p = 0.6400, ANCOVA; The ANCOVA model includes the fixed categorical effect of treatment and the continuous covariate of baseline LDL cholesterol; Mean Difference (Final Values) = 0.4, 95.47% CI 2-sided [-1.3 to 2.1], Standard Error of Mean 0.9 — Mean difference = Linagliptin mean - Glimepiride mean
Statistical Analysis 2: Comparison: Linagliptin vs Glimepiride; HDL cholesterol, this was the fifth step in a pre-defined hierarchical testing approach; Test type: Other; p = 0.0497, ANCOVA; The ANCOVA model includes the fixed categorical effect of treatment and the continuous covariate of baseline HDL cholesterol; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [0.0 to 1.0], Standard Error of Mean 0.2 — Mean difference = Linagliptin mean - Glimepiride mean
Statistical Analysis 3: Comparison: Linagliptin vs Glimepiride; Total cholesterol, this was the fifth step in a pre-defined hierarchical testing approach; Test type: Other; p = 0.6823, ANCOVA; The ANCOVA model includes the fixed categorical effect of treatment and the continuous covariate of baseline total cholesterol; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-2.4 to 1.6], Standard Error of Mean 1.0 — Mean difference = Linagliptin mean - Glimepiride mean

12. Secondary Outcome: Change From Baseline to Final Visit in Triglycerides
Description: Change from baseline to final visit in triglycerides is presented as secondary diabetes-related endpoint. Least square mean is adjusted mean. The Final Visit value referred to the last value obtained on-treatment.
Time Frame: Baseline and week 432
Population: TS w/o duplicates, participants on treatment
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 2788 | 2762
mg/dL | 1.7 (2.2) | 5.2 (2.2)
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; This was the fifth step in a pre-defined hierarchical testing approach; Test type: Other; p = 0.2678, ANCOVA; The ANCOVA model includes the fixed categorical effect of treatment and the continuous covariate of baseline FPG; Mean Difference (Final Values) = -3.5, 95% CI 2-sided [-9.6 to 2.7], Standard Error of Mean 3.1 — Mean difference = Linagliptin mean - Glimepiride mean

13. Secondary Outcome: Change From Baseline to Final Visit in Creatinine
Description: Change from baseline to final visit in creatinine is presented as secondary diabetes-related endpoint. Least square mean is adjusted mean. The Final Visit value referred to the last value obtained on-treatment.
Time Frame: Baseline and week 432
Population: TS w/o duplicates, participants on treatment
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 2917 | 2898
mg/dL | 0.08 (0.01) | 0.09 (0.01)
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; This was the fifth step in a pre-defined hierarchical testing approach; Test type: Other; p = 0.5165, ANCOVA; The ANCOVA model includes the fixed categorical effect of treatment and the continuous covariate of baseline creatinine; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.03 to 0.01], Standard Error of Mean 0.01 — Mean difference = Linagliptin mean - Glimepiride mean

14. Secondary Outcome: Change From Baseline to Final Visit in Estimated Glomerular Filtration Rate (eGFR)
Description: Change from baseline to final visit in eGFR is presented as secondary diabetes-related endpoint. Least square mean is adjusted mean. The Final Visit value referred to the last value obtained on-treatment.
Time Frame: Baseline and week 432
Population: TS w/o duplicates, participants on treatment
Measure: Least Squares Mean (Standard Error); unit: mL/minute/1.73 meter^2
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 2917 | 2898
mL/minute/1.73 meter^2 | -4.0 (0.3) | -5.0 (0.3)
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; This was the fifth step in a pre-defined hierarchical testing approach; Test type: Other; p = 0.5165, ANCOVA; The ANCOVA model includes the fixed categorical effect of treatment and the continuous covariate of baseline eGFR; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [0.2 to 1.8], Standard Error of Mean 0.4 — Mean difference = Linagliptin mean - Glimepiride mean

15. Secondary Outcome: Change From Baseline to Final Visit in Urine Albumin Creatinine Ratio (UACR)
Description: Change from baseline to final visit in UACR is presented as secondary diabetes-related endpoint. Least square mean is adjusted geometric mean (gMean) ratio. The Final Visit value referred to the last value obtained on-treatment.
Time Frame: Baseline and week 432
Population: TS w/o duplicates, participants on treatment
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/ gcrea
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 2904 | 2880
mg/ gcrea | 1.52 (1.83) | 1.57 (1.83)
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; This was the fifth step in a pre-defined hierarchical testing approach; Test type: Other; p = 0.2921, ANCOVA; The ANCOVA model includes the fixed categorical effect of treatment and the continuous covariate of baseline UACR; geometric mean (gMean) ratio (%) = 0.97, 95% CI 2-sided [0.91 to 1.03] — gMean ration= Linagliptin mean/ Glimepiride mean

16. Secondary Outcome: Percentage of Participants With Transition in Albuminuria Classes
Description: Percentage of patients with transition in albuminuria classes is presented as secondary endpoint. Data for last value on treatment (LVOT) to baseline (base) is presented.
Time Frame: Baseline and week 432
Population: TS w/o duplicates, participants on treatment
Measure: Number; unit: Percentage of participants (%)
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 3014 | 3000
Percentage of participants (%)
  Base (<30mg/gcrea) LVOT (<30mg/gcrea) | 58.4 | 57.7
  Base(<30mg/gcrea)LVOT(>=30 to<=300mg/gcrea) | 14.1 | 16.0
  Base (<30 mg/gcrea) LVOT (>300 mg/gcrea) | 1.4 | 1.4
  Base (>=30 to <=300 mg/gcrea) LVOT(<30mg/gcrea) | 5.4 | 5.1
  Base(>=30to<=300mg/gcrea)LVOT(>=30to<=300mg/gcrea) | 12.7 | 12.1
  Base (>=30 to <=300 mg/gcrea) LVOT(>300 mg/gcrea) | 3.5 | 3.7
  Base (>300 mg/gcrea) LVOT (<30 mg/gcrea) | 0.1 | 0.3
  Base (>300 mg/gcrea) LVOT(>=30 to<=300mg/gcrea) | 0.8 | 0.9
  Base (>300 mg/gcrea) LVOT(>300 mg/gcrea) | 3.4 | 2.7

17. Secondary Outcome: Change From Baseline of Insulin Secretion Rate (ISR) at Fixed Glucose Concentration at 208 Weeks
Description: The endpoint change from baseline of ISR at fixed glucose concentration at 208 weeks as derived from a 3-hour meal tolerance test is Beta-cell function sub-study endpoint.
Time Frame: Baseline and week 208
Population: Meal tolerance test(MTT) last observation carried forward(LOCF) set: Randomised and treated patients with one dose of study drug and signed the sub-study Informed Consent with valid baseline and on-treatment MTT. If values taken after rescue medication intake will be set to missing, last observed on-treatment value was carry forwarded.
Measure: Mean (Standard Error); unit: Picomol/ minute/meter^2 (pmol/min/m²)
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 40 | 48
Picomol/ minute/meter^2 (pmol/min/m²) | 11.07 (15.07) | 6.95 (13.76)
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; Test type: Equivalence — This was the fifth step in a pre-defined hierarchical testing approach; p = 0.8402, ANCOVA; The ANCOVA model includes the fixed categorical effects of treatment and the continuous covariate of baseline ISR; Mean Difference (Net) = 4.13, 95% CI 2-sided [-36.46 to 44.71] — Mean difference= Linagliptin mean- Glimepiride mean

18. Secondary Outcome: Percentage of Participants With Occurrence of Accelerated Cognitive Decline at End of Follow-up
Description: Occurrence of accelerated cognitive decline based on regression based index (RBI) score at end of follow-up (a dichotomous outcome measure; presence or absence of accelerated cognitive decline) is Cognition sub-study endpoint.
Time Frame: 433 weeks
Population: Full analysis set cognition(FAS-COG): Randomised and treated patients with one dose of study drug, baseline assessment (the z-scores, A&E or Mini-mental state examination(MMSE) can be calculated), years of formal education with baseline MMSE≥24 and at least one on-treatment assessment (of which at least one of the RBI scores can be calculated).
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 1618 | 1545
Percentage of participants (%) | 27.8 [25.6 to 30.0] | 27.6 [25.4 to 29.9]
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; This was the fifth step in a pre-defined hierarchical testing approach; Test type: Other; p = 0.9112, Regression, Logistic; Logistic regression model with terms for treatment as a fixed effect with Wald confidence Interval was used; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.86 to 1.18] — Linagliptin vs. Glimepiride odds is presented

19. Secondary Outcome: Continuous Glucose Monitoring (CGM) Sub-study: Change From Baseline in the Inter-quartile Range of Diurnal Glucose Variability (Milligrams/ Deciliter) to End of Study
Description: Baseline data for the continuous glucose monitoring sub-study was collected and analyzed. However, the participant number was far less than original planned. The study was stopped early around week 64 (V9) due to recruitment issues and data were not pre-specified to be analyzed and reported at week 64 time point as target was with an estimated time point of 432 weeks for primary or secondary end points. Thus this endpoint was not analysed and only the baseline data collected were analysed and the results are reported in this CGM substudy endpoint.
Time Frame: Baseline
Population: The sub-study was stopped early and required target with an estimated time point of 432 weeks was not achieved for this endpoint. Thus the data were not unblinded and only the baseline data collected were reported overall and not by treatment arm for this endpoint.
Measure: Mean (Standard Deviation); unit: Milligrams/ deciliter (mg/ dL)
Groups:
- All Participants: After 2-4 weeks placebo run-in phase, participants were administered 1 tablet of placebo matching linagliptin plus 1 over-encapsulated tablet of 1 to 4 mg glimepiride, which was uptitrated in 4-week intervals during the first 16 weeks of treatment to the next dose or 1 tablet of 5 milligram (mg) linagliptin plus 1 over-encapsulated tablet of placebo matching glimepiride, which was uptitrated in 4-week intervals during the first 16 weeks of treatment to the next dose. All doses were administered once daily orally up to an estimated 432 weeks treatment period.
Arm/Group | All Participants
Number analyzed (Participants) | 44
Milligrams/ deciliter (mg/ dL) | 44.2 (12.6)

20. Secondary Outcome: CGM Sub-study : Change From Baseline in the Inter-quartile Range of Diurnal Glucose Variability (Millimoles/ Litre) to End of Study
Description: as for outcome 19
Time Frame: Baseline
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Millimoles/ Litre (mmol/L)
Arm/Group | All Participants
Number analyzed (Participants) | 44
Millimoles/ Litre (mmol/L) | 2.45 (0.7)

ADVERSE EVENTS:
Time Frame: From start of the treatment until 7 days after the end of treatment, up to 433 weeks.
Arm/Group | Linagliptin | Glimepiride
All-Cause Mortality (participants affected / at risk) | 308/3023 | 336/3010
Serious Adverse Events (participants affected / at risk) | 1403/3023 | 1448/3010
Other Adverse Events (participants affected / at risk) | 2376/3023 | 2504/3010
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Linagliptin (N=3023) | Glimepiride (N=3010)
Anaemia (Blood and lymphatic system disorders) | 14 | 18
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 6 | 1
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 3
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 5 | 1
Splenic haematoma (Blood and lymphatic system disorders) | 1 | 0
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 18 | 12
Acute left ventricular failure (Cardiac disorders) | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 52 | 56
Adams-Stokes syndrome (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 37 | 40
Angina unstable (Cardiac disorders) | 54 | 65
Aortic valve disease (Cardiac disorders) | 1 | 2
Aortic valve incompetence (Cardiac disorders) | 1 | 1
Aortic valve stenosis (Cardiac disorders) | 5 | 4
Arrhythmia (Cardiac disorders) | 4 | 5
Arteriosclerosis coronary artery (Cardiac disorders) | 4 | 4
Atrial fibrillation (Cardiac disorders) | 39 | 48
Atrial flutter (Cardiac disorders) | 23 | 14
Atrial tachycardia (Cardiac disorders) | 2 | 2
Atrioventricular block (Cardiac disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 10 | 8
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 3 | 3
Bradyarrhythmia (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 6 | 7
Bundle branch block (Cardiac disorders) | 1 | 0
Bundle branch block left (Cardiac disorders) | 1 | 3
Cardiac aneurysm (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 4 | 8
Cardiac asthma (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 3 | 1
Cardiac failure (Cardiac disorders) | 58 | 53
Cardiac failure acute (Cardiac disorders) | 7 | 6
Cardiac failure chronic (Cardiac disorders) | 9 | 12
Cardiac failure congestive (Cardiac disorders) | 37 | 45
Cardiac perforation (Cardiac disorders) | 1 | 0
Cardiac valve disease (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 4 | 2
Cardiogenic shock (Cardiac disorders) | 2 | 4
Cardiomegaly (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 2
Cardiopulmonary failure (Cardiac disorders) | 1 | 1
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Conduction disorder (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 1 | 2
Cor pulmonale (Cardiac disorders) | 0 | 3
Coronary artery disease (Cardiac disorders) | 43 | 42
Coronary artery dissection (Cardiac disorders) | 1 | 0
Coronary artery insufficiency (Cardiac disorders) | 2 | 1
Coronary artery occlusion (Cardiac disorders) | 3 | 2
Coronary artery stenosis (Cardiac disorders) | 4 | 12
Diastolic dysfunction (Cardiac disorders) | 1 | 0
Extrasystoles (Cardiac disorders) | 0 | 1
Heart valve incompetence (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 4 | 2
Left ventricular dysfunction (Cardiac disorders) | 2 | 0
Left ventricular failure (Cardiac disorders) | 2 | 4
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0
Long QT syndrome (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 2
Mitral valve stenosis (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 49 | 64
Myocardial ischaemia (Cardiac disorders) | 14 | 9
Myocardial rupture (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 2 | 2
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 3
Postinfarction angina (Cardiac disorders) | 1 | 1
Prinzmetal angina (Cardiac disorders) | 1 | 1
Pulmonary valve stenosis (Cardiac disorders) | 0 | 1
Right ventricular dysfunction (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 1 | 1
Silent myocardial infarction (Cardiac disorders) | 5 | 5
Sinoatrial block (Cardiac disorders) | 1 | 0
Sinus arrest (Cardiac disorders) | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 1
Sinus node dysfunction (Cardiac disorders) | 4 | 5
Sinus tachycardia (Cardiac disorders) | 2 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 7
Tachyarrhythmia (Cardiac disorders) | 2 | 1
Tachycardia (Cardiac disorders) | 5 | 2
Tachycardia paroxysmal (Cardiac disorders) | 0 | 2
Thyrotoxic cardiomyopathy (Cardiac disorders) | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1
Trifascicular block (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 4 | 2
Ventricular fibrillation (Cardiac disorders) | 0 | 2
Ventricular hypokinesia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 4 | 1
Wolff-Parkinson-White syndrome (Cardiac disorders) | 1 | 0
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 0 | 1
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0
Choledochal cyst (Congenital, familial and genetic disorders) | 1 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1 | 0
Corneal dystrophy (Congenital, familial and genetic disorders) | 1 | 0
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 | 1
Exomphalos (Congenital, familial and genetic disorders) | 1 | 0
Fibrous dysplasia of bone (Congenital, familial and genetic disorders) | 1 | 0
Hereditary haemochromatosis (Congenital, familial and genetic disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 2 | 3
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 | 0
Ichthyosis (Congenital, familial and genetic disorders) | 0 | 1
Left ventricle outflow tract obstruction (Congenital, familial and genetic disorders) | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 3 | 6
Porokeratosis (Congenital, familial and genetic disorders) | 1 | 2
Stargardt's disease (Congenital, familial and genetic disorders) | 1 | 0
Urachal abnormality (Congenital, familial and genetic disorders) | 0 | 1
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 | 0
Aural polyp (Ear and labyrinth disorders) | 1 | 0
Conductive deafness (Ear and labyrinth disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 7 | 2
Deafness neurosensory (Ear and labyrinth disorders) | 3 | 6
Deafness unilateral (Ear and labyrinth disorders) | 0 | 4
Ear canal stenosis (Ear and labyrinth disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Inner ear disorder (Ear and labyrinth disorders) | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 1 | 0
Mixed deafness (Ear and labyrinth disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 9 | 12
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Basedow's disease (Endocrine disorders) | 1 | 0
Goitre (Endocrine disorders) | 3 | 4
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypoparathyroidism (Endocrine disorders) | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 1
Thyroid mass (Endocrine disorders) | 1 | 0
Age-related macular degeneration (Eye disorders) | 0 | 1
Amaurosis (Eye disorders) | 0 | 1
Amaurosis fugax (Eye disorders) | 2 | 3
Angle closure glaucoma (Eye disorders) | 4 | 1
Aphakia (Eye disorders) | 1 | 0
Blepharitis (Eye disorders) | 0 | 1
Blindness (Eye disorders) | 1 | 0
Blindness transient (Eye disorders) | 0 | 1
Blindness unilateral (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 16 | 21
Chalazion (Eye disorders) | 0 | 1
Detachment of retinal pigment epithelium (Eye disorders) | 0 | 1
Diabetic retinopathy (Eye disorders) | 1 | 2
Diplopia (Eye disorders) | 0 | 1
Dry age-related macular degeneration (Eye disorders) | 0 | 2
Endocrine ophthalmopathy (Eye disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 1 | 0
Eye swelling (Eye disorders) | 1 | 0
Eyelid ptosis (Eye disorders) | 1 | 2
Eyelid rash (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 29 | 31
Iris neovascularisation (Eye disorders) | 1 | 0
Keratitis (Eye disorders) | 0 | 1
Lens dislocation (Eye disorders) | 1 | 0
Macular degeneration (Eye disorders) | 12 | 11
Macular fibrosis (Eye disorders) | 5 | 6
Macular hole (Eye disorders) | 2 | 0
Neovascular age-related macular degeneration (Eye disorders) | 0 | 1
Open angle glaucoma (Eye disorders) | 0 | 1
Panophthalmitis (Eye disorders) | 2 | 0
Pterygium (Eye disorders) | 0 | 1
Retinal artery embolism (Eye disorders) | 2 | 1
Retinal artery occlusion (Eye disorders) | 3 | 0
Retinal degeneration (Eye disorders) | 2 | 0
Retinal detachment (Eye disorders) | 6 | 7
Retinal tear (Eye disorders) | 2 | 2
Retinal vein occlusion (Eye disorders) | 2 | 2
Retinopathy (Eye disorders) | 0 | 1
Ulcerative keratitis (Eye disorders) | 1 | 3
Uveitic glaucoma (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 1
Vitreous adhesions (Eye disorders) | 1 | 0
Vitreous degeneration (Eye disorders) | 0 | 1
Vitreous detachment (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 2 | 2
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 7 | 7
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 1
Acute abdomen (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 2
Appendiceal mucocoele (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 3
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 1
Bezoar (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 6 | 2
Colitis ischaemic (Gastrointestinal disorders) | 2 | 1
Colon dysplasia (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 3
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Dental necrosis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 5
Diverticulum (Gastrointestinal disorders) | 1 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 2
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 2 | 0
Duodenal polyp (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 3 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 4
Duodenitis (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 2
Enteritis (Gastrointestinal disorders) | 3 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1
Erosive duodenitis (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 4 | 3
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 3 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 5 | 6
Gastritis erosive (Gastrointestinal disorders) | 0 | 3
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 1
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 16 | 10
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 3
Haematochezia (Gastrointestinal disorders) | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 3 | 2
Hiatus hernia (Gastrointestinal disorders) | 1 | 2
Ileus (Gastrointestinal disorders) | 3 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 4
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 2
Inguinal hernia (Gastrointestinal disorders) | 18 | 14
Intestinal haematoma (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Intestinal mass (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 3 | 4
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Jejunal perforation (Gastrointestinal disorders) | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 6 | 9
Lip swelling (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 3
Lumbar hernia (Gastrointestinal disorders) | 1 | 0
Malignant bowel obstruction (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 3 | 4
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 5
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0
Oesophageal fistula (Gastrointestinal disorders) | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Pancreatic failure (Gastrointestinal disorders) | 1 | 0
Pancreatic mass (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 10 | 11
Pancreatitis acute (Gastrointestinal disorders) | 8 | 8
Pancreatitis chronic (Gastrointestinal disorders) | 5 | 2
Pancreatitis necrotising (Gastrointestinal disorders) | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1
Peptic ulcer perforation (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 2
Rectal polyp (Gastrointestinal disorders) | 1 | 0
Retroperitoneal fibrosis (Gastrointestinal disorders) | 1 | 0
Salivary gland calculus (Gastrointestinal disorders) | 1 | 0
Salivary gland mass (Gastrointestinal disorders) | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 5 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 1
Tongue oedema (Gastrointestinal disorders) | 0 | 1
Tongue ulceration (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 4 | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 | 4
Vomiting (Gastrointestinal disorders) | 3 | 4
Adhesion (General disorders) | 1 | 0
Adverse drug reaction (General disorders) | 1 | 0
Asthenia (General disorders) | 3 | 7
Cardiac death (General disorders) | 7 | 3
Chest discomfort (General disorders) | 3 | 6
Chest pain (General disorders) | 50 | 52
Chills (General disorders) | 0 | 1
Condition aggravated (General disorders) | 0 | 1
Death (General disorders) | 20 | 20
Discomfort (General disorders) | 1 | 0
Exercise tolerance decreased (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 3
Fibrosis (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 3 | 4
Hernia (General disorders) | 1 | 0
Hyperthermia (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Implant site extravasation (General disorders) | 1 | 0
Implant site haematoma (General disorders) | 0 | 1
Malaise (General disorders) | 3 | 2
Mass (General disorders) | 1 | 0
Multi-organ disorder (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 7
Non-cardiac chest pain (General disorders) | 8 | 8
Oedema peripheral (General disorders) | 2 | 1
Puncture site haemorrhage (General disorders) | 1 | 0
Pyrexia (General disorders) | 7 | 8
Retention cyst (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 3 | 1
Sudden death (General disorders) | 9 | 4
Swelling (General disorders) | 1 | 0
Vascular stent stenosis (General disorders) | 3 | 1
Acute hepatic failure (Hepatobiliary disorders) | 0 | 2
Bile duct obstruction (Hepatobiliary disorders) | 2 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 6 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 2 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 20 | 16
Cholecystitis acute (Hepatobiliary disorders) | 9 | 5
Cholecystitis chronic (Hepatobiliary disorders) | 3 | 0
Cholelithiasis (Hepatobiliary disorders) | 20 | 14
Cholestasis (Hepatobiliary disorders) | 0 | 1
Cholestatic liver injury (Hepatobiliary disorders) | 1 | 0
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 2 | 0
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0
Gallbladder necrosis (Hepatobiliary disorders) | 1 | 0
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 3 | 6
Hepatic cyst (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 1
Hepatic fibrosis (Hepatobiliary disorders) | 0 | 1
Hepatic lesion (Hepatobiliary disorders) | 0 | 1
Hepatic mass (Hepatobiliary disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 6 | 5
Hepatitis acute (Hepatobiliary disorders) | 2 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Hydrocholecystis (Hepatobiliary disorders) | 1 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 2 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 2 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 2
Allergy to vaccine (Immune system disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 2 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 1
Abscess (Infections and infestations) | 1 | 0
Abscess intestinal (Infections and infestations) | 1 | 0
Abscess jaw (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 3 | 3
Abscess neck (Infections and infestations) | 1 | 0
Acarodermatitis (Infections and infestations) | 0 | 1
Actinomycotic pulmonary infection (Infections and infestations) | 1 | 0
Acute hepatitis C (Infections and infestations) | 0 | 1
Administration site cellulitis (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 2
Appendiceal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 5 | 5
Appendicitis perforated (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 4
Arthritis infective (Infections and infestations) | 1 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 4 | 1
Bacterial sepsis (Infections and infestations) | 1 | 2
Biliary sepsis (Infections and infestations) | 0 | 1
Body tinea (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 15 | 11
Campylobacter gastroenteritis (Infections and infestations) | 1 | 1
Candida sepsis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 17 | 18
Cellulitis staphylococcal (Infections and infestations) | 0 | 1
Cholecystitis infective (Infections and infestations) | 1 | 1
Chronic tonsillitis (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0
Colon gangrene (Infections and infestations) | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Creutzfeldt-Jakob disease (Infections and infestations) | 0 | 2
Cystitis (Infections and infestations) | 0 | 3
Cystitis escherichia (Infections and infestations) | 0 | 1
Dengue fever (Infections and infestations) | 0 | 3
Device related infection (Infections and infestations) | 0 | 1
Device related sepsis (Infections and infestations) | 0 | 1
Diabetic foot infection (Infections and infestations) | 2 | 0
Diabetic gangrene (Infections and infestations) | 1 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 6 | 6
Empyema (Infections and infestations) | 0 | 2
Encephalitis (Infections and infestations) | 0 | 2
Endocarditis (Infections and infestations) | 1 | 1
Endocarditis bacterial (Infections and infestations) | 1 | 0
Enteritis infectious (Infections and infestations) | 2 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 2 | 2
Epiglottitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 3 | 11
Escherichia sepsis (Infections and infestations) | 1 | 0
External ear cellulitis (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 1 | 1
Fungal infection (Infections and infestations) | 1 | 0
Gallbladder abscess (Infections and infestations) | 2 | 1
Gangrene (Infections and infestations) | 3 | 4
Gastric ulcer helicobacter (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 17 | 17
Gastroenteritis clostridial (Infections and infestations) | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 2 | 0
Gastroenteritis viral (Infections and infestations) | 3 | 2
Gastrointestinal infection (Infections and infestations) | 1 | 0
Gingival abscess (Infections and infestations) | 1 | 0
Graft infection (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 2 | 0
Haematoma infection (Infections and infestations) | 1 | 1
Haemophilus infection (Infections and infestations) | 0 | 1
Helicobacter gastritis (Infections and infestations) | 2 | 1
Hepatitis A (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 1 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 9
Infected bite (Infections and infestations) | 1 | 0
Infected dermal cyst (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 2 | 0
Infection (Infections and infestations) | 1 | 3
Infectious colitis (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 0 | 2
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 | 1
Infective spondylitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 8
Intervertebral discitis (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 1 | 2
Localised infection (Infections and infestations) | 2 | 1
Lower respiratory tract infection (Infections and infestations) | 4 | 4
Lung infection (Infections and infestations) | 1 | 2
Lymphangitis (Infections and infestations) | 0 | 1
Mediastinitis (Infections and infestations) | 0 | 1
Medical device site infection (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Meningitis aseptic (Infections and infestations) | 0 | 1
Meningitis bacterial (Infections and infestations) | 1 | 1
Meningitis viral (Infections and infestations) | 1 | 0
Meningoencephalitis viral (Infections and infestations) | 0 | 1
Morganella infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2
Necrotising fasciitis (Infections and infestations) | 0 | 1
Nosocomial infection (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 0 | 2
Osteomyelitis (Infections and infestations) | 8 | 3
Osteomyelitis chronic (Infections and infestations) | 1 | 0
Osteomyelitis fungal (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Otitis media chronic (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 1 | 0
Perichondritis (Infections and infestations) | 0 | 1
Periodontitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 83 | 83
Pneumonia bacterial (Infections and infestations) | 3 | 0
Pneumonia necrotising (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 2 | 0
Pneumonia viral (Infections and infestations) | 0 | 1
Post procedural cellulitis (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 1 | 3
Postoperative abscess (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 3 | 4
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Purulence (Infections and infestations) | 0 | 1
Pyelitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 8 | 4
Pyelonephritis acute (Infections and infestations) | 4 | 2
Pyelonephritis fungal (Infections and infestations) | 1 | 0
Pyonephrosis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 2 | 7
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Retroperitoneal abscess (Infections and infestations) | 0 | 1
Rotavirus infection (Infections and infestations) | 0 | 1
Salmonellosis (Infections and infestations) | 0 | 1
Scrotal abscess (Infections and infestations) | 0 | 1
Scrub typhus (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 17 | 24
Septic arthritis streptococcal (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 6 | 7
Sialoadenitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1
Small intestine gangrene (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 2
Staphylococcal infection (Infections and infestations) | 1 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 2
Tooth infection (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 3
Ureteritis (Infections and infestations) | 2 | 0
Urethritis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 30 | 31
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1
Urinary tract infection fungal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 7 | 6
Varicella (Infections and infestations) | 0 | 1
Vestibular neuronitis (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 1 | 2
Vulval abscess (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 2 | 4
Accident (Injury, poisoning and procedural complications) | 1 | 3
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1
Anaesthetic complication cardiac (Injury, poisoning and procedural complications) | 0 | 1
Anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 6 | 11
Arterial restenosis (Injury, poisoning and procedural complications) | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 0 | 1
Bladder injury (Injury, poisoning and procedural complications) | 1 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1
Bone fragmentation (Injury, poisoning and procedural complications) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 2 | 1
Brain herniation (Injury, poisoning and procedural complications) | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 1
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 | 1
Carotid artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0
Chemical burn (Injury, poisoning and procedural complications) | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 3
Conjunctival laceration (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 4 | 5
Coronary artery reocclusion (Injury, poisoning and procedural complications) | 0 | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 3
Craniocerebral injury (Injury, poisoning and procedural complications) | 5 | 1
Crush injury (Injury, poisoning and procedural complications) | 0 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Eye contusion (Injury, poisoning and procedural complications) | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 2
Fall (Injury, poisoning and procedural complications) | 31 | 44
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 | 4
Femur fracture (Injury, poisoning and procedural complications) | 9 | 6
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 2
Foot fracture (Injury, poisoning and procedural complications) | 1 | 4
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 3
Fracture of penis (Injury, poisoning and procedural complications) | 1 | 0
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 2 | 2
Head injury (Injury, poisoning and procedural complications) | 5 | 4
Hip fracture (Injury, poisoning and procedural complications) | 7 | 16
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 6
Ilium fracture (Injury, poisoning and procedural complications) | 1 | 0
Impacted fracture (Injury, poisoning and procedural complications) | 1 | 1
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 3 | 1
Inflammation of wound (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Injury corneal (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 6 | 6
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 5 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 4
Limb injury (Injury, poisoning and procedural complications) | 2 | 3
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 7 | 5
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3 | 2
Meniscus injury (Injury, poisoning and procedural complications) | 6 | 4
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 2
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 4 | 1
Patella fracture (Injury, poisoning and procedural complications) | 2 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Pneumoconiosis (Injury, poisoning and procedural complications) | 0 | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 | 0
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 | 1
Post procedural urine leak (Injury, poisoning and procedural complications) | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Postoperative renal failure (Injury, poisoning and procedural complications) | 0 | 1
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 2 | 1
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 2 | 6
Rib fracture (Injury, poisoning and procedural complications) | 5 | 4
Road traffic accident (Injury, poisoning and procedural complications) | 13 | 7
Scar (Injury, poisoning and procedural complications) | 0 | 1
Shunt occlusion (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 8 | 1
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 4
Splenic injury (Injury, poisoning and procedural complications) | 1 | 0
Stab wound (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 5 | 5
Subdural haematoma (Injury, poisoning and procedural complications) | 5 | 7
Subdural haemorrhage (Injury, poisoning and procedural complications) | 5 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 6 | 3
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 3 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 2
Transplant dysfunction (Injury, poisoning and procedural complications) | 0 | 1
Traumatic arthritis (Injury, poisoning and procedural complications) | 1 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 3
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 2
Urethral injury (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 2 | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 0
Wound necrosis (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase increased (Investigations) | 6 | 7
Amylase increased (Investigations) | 3 | 0
Anticoagulation drug level below therapeutic (Investigations) | 0 | 1
Arteriogram coronary (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 6 | 7
Blood alkaline phosphatase increased (Investigations) | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatine phosphokinase MB increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 12 | 11
Blood pressure decreased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Body temperature increased (Investigations) | 1 | 0
Cardiac stress test abnormal (Investigations) | 1 | 0
Computerised tomogram head abnormal (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 2 | 0
Electrocardiogram ST segment depression (Investigations) | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 2 | 2
Electrocardiogram abnormal (Investigations) | 1 | 0
Electrocardiogram ambulatory abnormal (Investigations) | 1 | 0
Full blood count decreased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 7 | 7
Glomerular filtration rate decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 2
Heart rate decreased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 2 | 1
Hepatitis C virus test (Investigations) | 1 | 0
International normalised ratio decreased (Investigations) | 1 | 1
International normalised ratio increased (Investigations) | 3 | 0
Lipase increased (Investigations) | 3 | 1
Liver function test abnormal (Investigations) | 0 | 2
Liver function test increased (Investigations) | 1 | 1
Myelocyte count increased (Investigations) | 0 | 1
Positron emission tomogram abnormal (Investigations) | 0 | 1
Prostatic specific antigen increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 4 | 1
Urine albumin/creatinine ratio increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 1
Weight increased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 13 | 10
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 3
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 2
Fluid overload (Metabolism and nutrition disorders) | 2 | 2
Gout (Metabolism and nutrition disorders) | 4 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 8
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 7 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 29
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 4
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 4 | 1
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 9
Arthritis (Musculoskeletal and connective tissue disorders) | 6 | 4
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 8
Bone atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 3 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 4 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 3
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 8 | 12
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1
Limb deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 11 | 7
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 49 | 63
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 9 | 13
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 4 | 3
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 7 | 5
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 4 | 12
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 8
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 3 | 2
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 7
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 39 | 33
Basosquamous carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 8
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 8
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 9
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 5
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Conjunctival melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cutaneous lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Enchondromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Ependymoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypopharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lentigo maligna recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 8
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 6
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 2
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Mucinous adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Myxofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 9
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Paranasal sinus and nasal cavity malignant neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 6
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pleural sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Porocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prolactin-producing pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 28 | 29
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Prostate cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Refractory anaemia with ringed sideroblasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 6
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Sebaceous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Skin angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Soft tissue sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 6
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 16
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of the hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Vipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 2 | 1
Aphasia (Nervous system disorders) | 1 | 1
Balance disorder (Nervous system disorders) | 0 | 1
Basal ganglia haematoma (Nervous system disorders) | 1 | 0
Basal ganglia haemorrhage (Nervous system disorders) | 2 | 0
Basal ganglia infarction (Nervous system disorders) | 2 | 1
Basilar artery stenosis (Nervous system disorders) | 0 | 1
Basilar artery thrombosis (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 1
Brain stem stroke (Nervous system disorders) | 0 | 2
Carotid artery aneurysm (Nervous system disorders) | 1 | 1
Carotid artery occlusion (Nervous system disorders) | 5 | 3
Carotid artery stenosis (Nervous system disorders) | 13 | 10
Carpal tunnel syndrome (Nervous system disorders) | 1 | 1
Central pain syndrome (Nervous system disorders) | 1 | 0
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0
Cerebellar infarction (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 3
Cerebral infarction (Nervous system disorders) | 14 | 13
Cerebral ischaemia (Nervous system disorders) | 3 | 1
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 51 | 61
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 1 | 1
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 2
Coma (Nervous system disorders) | 0 | 1
Coordination abnormal (Nervous system disorders) | 0 | 2
Dementia (Nervous system disorders) | 13 | 19
Dementia Alzheimer's type (Nervous system disorders) | 1 | 2
Diabetic neuropathy (Nervous system disorders) | 0 | 3
Dizziness (Nervous system disorders) | 11 | 7
Drop attacks (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 1
Encephalomalacia (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 4 | 11
Facial paresis (Nervous system disorders) | 0 | 1
Generalised non-convulsive epilepsy (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 2 | 1
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 6 | 3
Headache (Nervous system disorders) | 3 | 2
Hemianopia (Nervous system disorders) | 1 | 0
Hemianopia homonymous (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 6 | 4
Hemiplegia (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Hypertensive cerebrovascular disease (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 2
IIIrd nerve paralysis (Nervous system disorders) | 0 | 1
Internal carotid artery kinking (Nervous system disorders) | 0 | 2
Intracranial aneurysm (Nervous system disorders) | 1 | 2
Intracranial haematoma (Nervous system disorders) | 0 | 1
Intracranial mass (Nervous system disorders) | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 22 | 20
Lacunar infarction (Nervous system disorders) | 4 | 4
Lacunar stroke (Nervous system disorders) | 2 | 3
Loss of consciousness (Nervous system disorders) | 1 | 3
Lumbar radiculopathy (Nervous system disorders) | 1 | 2
Memory impairment (Nervous system disorders) | 1 | 1
Mental impairment (Nervous system disorders) | 1 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 2
Mononeuritis (Nervous system disorders) | 0 | 1
Monoparesis (Nervous system disorders) | 0 | 1
Myelopathy (Nervous system disorders) | 1 | 1
Neurological symptom (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Paralysis recurrent laryngeal nerve (Nervous system disorders) | 0 | 1
Paraparesis (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 1 | 2
Parkinsonism (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 5 | 5
Quadriplegia (Nervous system disorders) | 0 | 1
Radicular syndrome (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 2
Retinal migraine (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 7 | 7
Seizure (Nervous system disorders) | 6 | 6
Sensory disturbance (Nervous system disorders) | 0 | 1
Spinal claudication (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 1
Spinal cord disorder (Nervous system disorders) | 0 | 1
Spondylitic myelopathy (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 1
Subdural hygroma (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 17 | 18
Tension headache (Nervous system disorders) | 1 | 1
Thrombotic cerebral infarction (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 31 | 33
Tunnel vision (Nervous system disorders) | 1 | 0
Vascular dementia (Nervous system disorders) | 2 | 1
Vascular encephalopathy (Nervous system disorders) | 1 | 1
Vertebral artery aneurysm (Nervous system disorders) | 0 | 1
Vertebral artery stenosis (Nervous system disorders) | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 2 | 1
Device battery issue (Product Issues) | 1 | 1
Device defective (Product Issues) | 1 | 0
Device dislocation (Product Issues) | 1 | 3
Device failure (Product Issues) | 1 | 0
Device fastener issue (Product Issues) | 1 | 0
Device leakage (Product Issues) | 0 | 1
Device loosening (Product Issues) | 1 | 0
Device malfunction (Product Issues) | 2 | 0
Device occlusion (Product Issues) | 1 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0
Agitated depression (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 4 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 1
Burnout syndrome (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 3
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 6 | 4
Delirium tremens (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 3 | 6
Depression suicidal (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 2 | 0
Encopresis (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 5
Mental disorder (Psychiatric disorders) | 2 | 1
Mental status changes (Psychiatric disorders) | 2 | 5
Panic attack (Psychiatric disorders) | 0 | 1
Panic disorder (Psychiatric disorders) | 1 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 1 | 0
Somatic symptom disorder (Psychiatric disorders) | 1 | 2
Substance abuse (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 3 | 1
Suicide attempt (Psychiatric disorders) | 1 | 1
Transient psychosis (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 47 | 41
Anuria (Renal and urinary disorders) | 0 | 1
Atonic urinary bladder (Renal and urinary disorders) | 0 | 1
Bladder neck obstruction (Renal and urinary disorders) | 0 | 1
Bladder outlet obstruction (Renal and urinary disorders) | 1 | 1
Bladder perforation (Renal and urinary disorders) | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 1 | 2
Calculus bladder (Renal and urinary disorders) | 1 | 2
Calculus urinary (Renal and urinary disorders) | 2 | 0
Chronic kidney disease (Renal and urinary disorders) | 15 | 6
Diabetic nephropathy (Renal and urinary disorders) | 1 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
End stage renal disease (Renal and urinary disorders) | 1 | 3
Glomerulonephritis (Renal and urinary disorders) | 0 | 1
Glomerulonephritis membranous (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 7 | 4
Hydronephrosis (Renal and urinary disorders) | 7 | 6
Hypertonic bladder (Renal and urinary disorders) | 0 | 1
Leukocyturia (Renal and urinary disorders) | 1 | 0
Lower urinary tract symptoms (Renal and urinary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 14 | 4
Nephrotic syndrome (Renal and urinary disorders) | 1 | 1
Obstructive nephropathy (Renal and urinary disorders) | 1 | 0
Prerenal failure (Renal and urinary disorders) | 1 | 1
Proteinuria (Renal and urinary disorders) | 1 | 1
Renal artery arteriosclerosis (Renal and urinary disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 3 | 1
Renal cyst (Renal and urinary disorders) | 0 | 2
Renal failure (Renal and urinary disorders) | 20 | 13
Renal impairment (Renal and urinary disorders) | 8 | 10
Renal mass (Renal and urinary disorders) | 1 | 0
Stag horn calculus (Renal and urinary disorders) | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0
Ureteral disorder (Renal and urinary disorders) | 1 | 0
Ureteral polyp (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 5 | 8
Urethral meatus stenosis (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 3 | 0
Urinary bladder polyp (Renal and urinary disorders) | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 13 | 3
Urinary tract obstruction (Renal and urinary disorders) | 0 | 2
Acquired phimosis (Reproductive system and breast disorders) | 0 | 1
Adenomyosis (Reproductive system and breast disorders) | 1 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 5 | 19
Breast pain (Reproductive system and breast disorders) | 0 | 1
Cystocele (Reproductive system and breast disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 1
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Ovarian disorder (Reproductive system and breast disorders) | 1 | 0
Pelvic prolapse (Reproductive system and breast disorders) | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Prostatic disorder (Reproductive system and breast disorders) | 1 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 1 | 0
Prostatism (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Rectocele (Reproductive system and breast disorders) | 1 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 4 | 4
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 2 | 4
Vulvar dysplasia (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 10
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 23 | 26
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Diaphragm muscle weakness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 22
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 16
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 6 | 11
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 14
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 2 | 4
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 2 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 4 | 3
Diabetic neuropathic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 3 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 1
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 3 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 4
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 4
Skin plaque (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 6
Solar lentigo (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0
Umbilical haematoma (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Loss of personal independence in daily activities (Social circumstances) | 1 | 1
Sexual abuse (Social circumstances) | 1 | 0
Cardiac operation (Surgical and medical procedures) | 1 | 0
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 1
Colostomy (Surgical and medical procedures) | 0 | 1
Colostomy closure (Surgical and medical procedures) | 1 | 0
Coronary arterial stent insertion (Surgical and medical procedures) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Implantable defibrillator insertion (Surgical and medical procedures) | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 3 | 3
Mitral valve replacement (Surgical and medical procedures) | 1 | 0
Prostatic operation (Surgical and medical procedures) | 1 | 0
Shoulder arthroplasty (Surgical and medical procedures) | 1 | 0
Spinal decompression (Surgical and medical procedures) | 1 | 0
Stent placement (Surgical and medical procedures) | 1 | 0
Thyroidectomy (Surgical and medical procedures) | 0 | 1
Transurethral prostatectomy (Surgical and medical procedures) | 0 | 1
Accelerated hypertension (Vascular disorders) | 1 | 0
Aneurysm (Vascular disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 5 | 7
Aortic aneurysm rupture (Vascular disorders) | 2 | 1
Aortic arteriosclerosis (Vascular disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 1 | 0
Aortic occlusion (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 3 | 3
Arterial occlusive disease (Vascular disorders) | 1 | 3
Arteriosclerosis (Vascular disorders) | 0 | 2
Arteritis (Vascular disorders) | 1 | 2
Atherosclerotic plaque rupture (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 4 | 6
Deep vein thrombosis (Vascular disorders) | 9 | 17
Diabetic vascular disorder (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 0 | 1
Embolism venous (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 1 | 0
Femoral artery aneurysm (Vascular disorders) | 1 | 0
Femoral artery embolism (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 4 | 3
Haemodynamic instability (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 12 | 9
Hypertensive crisis (Vascular disorders) | 15 | 21
Hypertensive emergency (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 5 | 3
Hypovolaemic shock (Vascular disorders) | 1 | 2
Infarction (Vascular disorders) | 0 | 2
Intermittent claudication (Vascular disorders) | 1 | 4
Ischaemia (Vascular disorders) | 1 | 2
Ischaemic limb pain (Vascular disorders) | 0 | 1
Lymphocele (Vascular disorders) | 2 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 6 | 12
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 10 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 1 | 2
Peripheral ischaemia (Vascular disorders) | 0 | 5
Peripheral vascular disorder (Vascular disorders) | 3 | 4
Shock (Vascular disorders) | 3 | 2
Thrombophlebitis (Vascular disorders) | 1 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 1 | 2
Venous thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Linagliptin (N=3023) | Glimepiride (N=3010)
Anaemia (Blood and lymphatic system disorders) | 208 | 178
Cataract (Eye disorders) | 219 | 203
Constipation (Gastrointestinal disorders) | 195 | 173
Diarrhoea (Gastrointestinal disorders) | 365 | 324
Nausea (Gastrointestinal disorders) | 157 | 164
Fatigue (General disorders) | 118 | 162
Oedema peripheral (General disorders) | 150 | 194
Bronchitis (Infections and infestations) | 315 | 340
Influenza (Infections and infestations) | 268 | 243
Nasopharyngitis (Infections and infestations) | 530 | 517
Upper respiratory tract infection (Infections and infestations) | 313 | 319
Urinary tract infection (Infections and infestations) | 318 | 312
Fall (Injury, poisoning and procedural complications) | 151 | 170
Lipase increased (Investigations) | 209 | 154
Hyperglycaemia (Metabolism and nutrition disorders) | 422 | 483
Hypoglycaemia (Metabolism and nutrition disorders) | 299 | 1067
Arthralgia (Musculoskeletal and connective tissue disorders) | 310 | 308
Back pain (Musculoskeletal and connective tissue disorders) | 388 | 368
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 150 | 181
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 224 | 261
Pain in extremity (Musculoskeletal and connective tissue disorders) | 215 | 224
Dizziness (Nervous system disorders) | 283 | 358
Headache (Nervous system disorders) | 268 | 295
Cough (Respiratory, thoracic and mediastinal disorders) | 284 | 290
Hypertension (Vascular disorders) | 430 | 452

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-04-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT01243424/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT01243424/SAP_001.pdf